CLINICAL TRIAL: NCT00658359
Title: A Phase 2, Multicenter, Open-label, Active Comparator-controlled, Extension Trial To Evaluate The Long-term Safety And Efficacy Of Cp-690,550 In Renal Allograft Recipients
Brief Title: Extension Study Of Subjects From Study A3921030 For The Prevention Of Acute Rejection In Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3921050; 2008-002345-23 (EudraCT Number)
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression; JAK inhibitor; kidney transplantation
MeSH Terms: interventions — Cyclosporine; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Arm 1 (Active Comparator): Treatment Arm 1 will also receive standard of care medications
  Interventions: Drug: Cyclosporine
- Treatment Arm 2 (Experimental): Treatment Arm 2 will also receive standard of care medications
  Interventions: Drug: CP-690,550
- Treatment Arm 3 (Experimental): Treatment Arm 3 will also receive standard of care medications
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Cyclosporine — Standard of care
  Arms: Treatment Arm 1
Drug: CP-690,550 — CP-690,550 tablets dosed BID Months 12-72
  Arms: Treatment Arm 2
Drug: CP-690,550 — CP-690,550 tablets dosed BID Months 12-72
  Arms: Treatment Arm 3

SUMMARY:
This is a study that will follow transplant patients from Study A3921030 to monitor for long term safety, tolerability and efficacy for 5 additional years, except in Portugal where the study will follow transplant patients through Month 36 posttransplant. Patients will continue their study medications that were previously assigned.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who successfully completed Study A3921030

Exclusion Criteria:

* Subjects who are on the waiting list for a second kidney transplant or any non-renal organ transplants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (65):
- United States (37):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai MedicalCenter, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford School of Medicine, Palo Alto, California
  - Stanford University Medical Center, Palo Alto, California
  - Balboa Institute of Transplantation, San Diego, California
  - California Institute of Renal Research, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center - Pacific Campus, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF Medical Center - Long Hospital, San Francisco, California
  - USCF Medical Center - Connie Frank Transplant Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Yale Physicians Building, New Haven, Connecticut
  - University Of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - NUCATS's Clinical Research Unit, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Investigational Drug Services (IDS) / UNC Healthcare, Chapel Hill, North Carolina
  - Transplant Clinic/UNC Heathcare, Chapel Hill, North Carolina
  - UNC Department of Surgery, Clinical Trials Consortium, Chapel Hill, North Carolina
  - UNC Department of Surgery/Abdominal Transplant Division, Chapel Hill, North Carolina
  - Division of Pharmacotherapy, School of Pharmacy, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina, Department of Medicine/Nephrology, Chapel Hill, North Carolina
  - Drexel University College of Medicine - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Department of Transplantation Surgery, Charleston, South Carolina
  - Nephrology Clinic, Charleston, South Carolina
  - Dallas Transplant Institute, Dallas, Texas
  - Annette C. and Harold C. Simmons Transplant Institute at Baylor University Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Department of Renal Medicine, Westmead, New South Wales
  - Central Northern Adelaide Renal and Transplantation Service, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (2):
  - Hopital Erasme, Anderlecht, Brussels Capital
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Brazil (4):
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital do Rim e Hipertensao, São Paulo, São Paulo
  - Ambulatorio Pos Transplante do Hospital do Rim a Hipertensao, São Paulo, São Paulo
  - Hospital do Rim e Hipertensao, São Paulo
- University of Alberta Hospital, Edmonton, Alberta, Canada
- Institut Klinicke a Experimentalni Mediciny, Praha 4 Krc, Czechia
- France (2):
  - Hopital Necker, Paris
  - CHRU de Nancy-Brabois - Service de Nephrologie, Vandœuvre-lès-Nancy
- Charite - Universitatsmedizin Berlin, Berlin, Germany
- Italy (2):
  - Istituto di Clinica Chirurgica, Universita Cattolica del Sacro Cuore, Roma, RM
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola Malpighi, Bologna
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Oslo universitetssykehus HF- Rikshospitalet, Oslo, Norway
- Akademicki Szpital Kliniczny im. J. Mikulicza - Radeckiego we Wroclawiu, Wroclaw, Poland
- Portugal (2):
  - Hospitais da Universidade de Coimbra, EPE, Coimbra
  - Hospital Curry Cabral, Lisbon
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Department of Surgery, Yonsei University College of Medicine Severance Hospital, Seoul
  - Asan Medical Center, Department of Surgery, Seoul
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921050&StudyName=Extension%20Study%20Of%20Subjects%20From%20Study%20A3921030%20For%20The%20Prevention%20Of%20Acute%20Rejection%20In%20Kidney%20Transplant%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and studied between 18 August 2008 and 18 February 2015. Those with 6-month time-weighted concentrations at 2-hours postdose (TWC2) above the median (Amendment 3), negative/unknown Epstein-Barr virus (EBV) at transplant, cytomegalovirus disease or lymphocyte-depleting agents posttransplant (Amendment 4) were discontinued
Pre-assignment Details: Participants who had completed 12 months treatment with tofacitinib or cyclosporine (CsA) in previous parent study (A3921030) continued study drugs for an additional 60 months in this extension study.
Groups:
- Cyclosporine: CsA was administered for up to 60 months as CsA microemulsion (Neoral® brand in the United States) orally twice daily (BID) in 2 equal doses approximately 12 hours apart. The dosage was adjusted to achieve a 12 hour trough whole blood level of approximately 75 to 200 nanograms per milliliter (ng/mL). Participants also received oral mycophenolate mofetil (MMF) 1 to 2 gram tablet daily throughout this extension study (or up to 3 mg daily for Black participants). Prednisone 5mg daily (or equivalent) was also maintained through at least 12 months posttransplant (parent study).
- Tofacitinib Less Intensive (LI): Tofacitinib was administered for up to 60 months. During the parent study (A3921030), participants received 15 milligram (mg) tablet orally BID for Months 1 to 3 posttransplant then 10 mg tablet orally BID from Month 4. On entry to this extension study (Month 12), the dose was continued and tapered to 5 mg BID as early as Month 12 and by Month 18 posttransplant. Total tofacitinib LI treatment was up to 72 months posttransplant (12 months parent study and 60 months extension). Participants also received oral MMF 1 to 2 gram tablet daily throughout this extension study. Prednisone 5mg daily (or equivalent) was also maintained through at least 12 months posttransplant (parent study).
- Tofacitinib More Intensive (MI): Tofacitinib was administered for up to 60 months. During the parent study (A3921030), participants received 15 mg tablet orally BID for Months 1 to 6 posttransplant then 10 mg tablet orally BID from Month 7. On entry to this extension study (Month 12), the dose was continued and tapered to 5 mg BID as early as Month 12 and by Month 18 posttransplant. Total tofacitinib MI treatment was up to 72 months posttransplant (12 months parent study and 60 months extension). Participants also received oral MMF 1 to 2 gram tablet daily throughout this extension study. Prednisone 5mg daily (or equivalent) was also maintained through at least 12 months posttransplant (parent study).
Period: Overall Study
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Started | 64 | 60 | 54
Completed | 36 | 15 | 8
Not Completed | 28 | 45 | 46
Not completed — Death | 3 | 1 | 2
Not completed — Adverse Event | 13 | 6 | 9
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Includes protocol Amendments 3 and 4 | 2 | 31 | 29
Not completed — Withdrawal by Subject | 7 | 4 | 2
Not completed — Lost to Follow-up | 2 | 2 | 4
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as those participants who received at least 1 dose of study drug in Study A3921050.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI) | Total
Number analyzed (Participants) | 64 | 60 | 54 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (12.7) | 45.7 (12.6) | 48.5 (10.9) | 46.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 14 | 53
  Male | 44 | 41 | 40 | 125

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Clinically Significant Infection by Visit
Description: Clinically significant infection was defined as the presence of documented infection confirmed by culture, biopsy, genomic, or serologic findings post-randomization and requiring hospitalization or parenteral anti-infective treatment, or otherwise deemed significant by the investigator. The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 61 | 55 | 52
Percentage of Participants
  Month 12 | 4.69 [2.46 to 6.91] | 8.33 [5.33 to 11.34] | 3.70 [1.54 to 5.87]
  Month 15 (n=59,54,44) | 7.81 [4.99 to 10.64] | 10.00 [6.74 to 13.26] | 18.52 [14.07 to 22.97]
  Month 18 (n=57,52,41) | 9.40 [6.33 to 12.48] | 13.33 [9.64 to 17.03] | 20.46 [15.83 to 25.09]
  Month 24 (n=54,48,34) | 11.02 [7.71 to 14.33] | 18.33 [14.13 to 22.54] | 24.49 [19.51 to 29.47]
  Month 30 (n=49,34,23) | 12.80 [9.23 to 16.36] | 25.42 [20.64 to 30.21] | 29.46 [24.00 to 34.92]
  Month 36 (n=46,28,12) | 14.62 [10.81 to 18.42] | 27.83 [22.79 to 32.87] | 34.89 [28.20 to 41.57]
  Month 42 (n=40,28,11) | 14.62 [10.81 to 18.42] | 27.83 [22.79 to 32.87] | 34.89 [28.20 to 41.57]
  Month 48 (n=37,28,11) | 16.81 [12.68 to 20.93] | 27.83 [22.79 to 32.87] | 34.89 [28.20 to 41.57]
  Month 54 (n=36,25,10) | 19.05 [14.62 to 23.48] | 33.08 [27.52 to 38.64] | 34.89 [28.20 to 41.57]
  Month 60 (n=34,21,10) | 19.05 [14.62 to 23.48] | 36.13 [30.26 to 41.99] | 34.89 [28.20 to 41.57]
  Month 66 (n=29,19,8) | 19.05 [14.62 to 23.48] | 36.13 [30.26 to 41.99] | 34.89 [28.20 to 41.57]
  Month 72 (n=24,15,7) | 21.94 [17.05 to 26.84] | 40.12 [33.73 to 46.51] | 43.03 [34.35 to 51.70]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.6694, Wald Test; Estimated rate difference = 2.19, 60% CI 2-sided [-2.12 to 6.50], Standard Error of Mean 5.12 — Tofacitinib LI minus CsA. Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.0873, Wald Test; Estimated rate difference = 10.71, 60% CI 2-sided [5.44 to 15.98], Standard Error of Mean 6.26 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.4912, Wald Test; Estimated rate difference = 3.93, 60% CI 2-sided [-0.87 to 8.74], Standard Error of Mean 5.71 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.0942, Wald Test; Estimated rate difference = 11.06, 60% CI 2-sided [5.50 to 16.62], Standard Error of Mean 6.61 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.2499, Wald Test; Estimated rate difference = 7.31, 60% CI 2-sided [1.96 to 12.66], Standard Error of Mean 6.36 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.0580, Wald Test; Estimated rate difference = 13.47, 60% CI 2-sided [7.49 to 19.45], Standard Error of Mean 7.10 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.0750, Wald Test; Estimated rate difference = 12.62, 60% CI 2-sided [6.66 to 18.59], Standard Error of Mean 7.09 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.0316, Wald Test; Estimated rate difference = 16.66, 60% CI 2-sided [10.14 to 23.19], Standard Error of Mean 7.75 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.0783, Wald Test; Estimated rate difference = 13.21, 60% CI 2-sided [6.90 to 19.53], Standard Error of Mean 7.50 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.0266, Wald Test; Estimated rate difference = 20.27, 60% CI 2-sided [12.58 to 27.96], Standard Error of Mean 9.14 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0783, Wald Test; Estimated rate difference = 13.21, 60% CI 2-sided [6.90 to 19.53], Standard Error of Mean 7.50 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.0266, Wald Test; Estimated rate difference = 20.27, 60% CI 2-sided [12.58 to 27.96], Standard Error of Mean 9.14 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.1545, Wald Test; Estimated rate difference = 11.02, 60% CI 2-sided [4.51 to 17.54], Standard Error of Mean 7.74 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.0528, Wald Test; Estimated rate difference = 18.08, 60% CI 2-sided [10.22 to 25.94], Standard Error of Mean 9.34 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0968, Wald Test; Estimated rate difference = 14.03, 60% CI 2-sided [6.92 to 21.14], Standard Error of Mean 8.45 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.0966, Wald Test; Estimated rate difference = 15.83, 60% CI 2-sided [7.81 to 23.85], Standard Error of Mean 9.53 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0507, Wald Test; Estimated rate difference = 17.07, 60% CI 2-sided [9.72 to 24.42], Standard Error of Mean 8.74 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.0966, Wald Test; Estimated rate difference = 15.83, 60% CI 2-sided [7.81 to 23.85], Standard Error of Mean 9.53 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0507, Wald Test; Estimated rate difference = 17.07, 60% CI 2-sided [9.72 to 24.42], Standard Error of Mean 8.74 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.0966, Wald Test; Estimated rate difference = 15.83, 60% CI 2-sided [7.81 to 23.85], Standard Error of Mean 9.53 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0574, Wald Test; Estimated rate difference = 18.17, 60% CI 2-sided [10.12 to 26.22], Standard Error of Mean 9.56 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.0749, Wald Test; Estimated rate difference = 21.08, 60% CI 2-sided [11.12 to 31.04], Standard Error of Mean 11.84 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 12; Test type: Superiority or Other; p = 0.4116, Wald Test; Estimated rate difference = 3.65, 60% CI 2-sided [-0.09 to 7.38], Standard Error of Mean 4.44 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 12; Test type: Superiority or Other; p = 0.7895, Wald Test; Estimated rate difference = -0.98, 60% CI 2-sided [-4.09 to 2.12], Standard Error of Mean 3.69 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference

2. Primary Outcome: Percentage of Participants With Malignancies
Description: All treatment-emergent malignancies in Study A3921050 were included as collected on the Malignancy Case Report Form page.
Time Frame: Months 12 through 72.
Population: Safety Analysis Set. Percentages use n (the number of participants with malignancies: 7,8,8 respectively) and include 1 participant in CsA and 2 in Tofacitinib LI from before dose reduction to 5 mg by Month 18 was implemented (protocol Amendment 1)
Measure: Number; unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 64 | 60 | 54
Percentage of Participants | 10.9 | 13.3 | 14.8
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Test type: Superiority or Other; p = 0.683, Chi-squared; Estimated rate difference = 2.4, 95% CI 2-sided [-9.1 to 13.9], Standard Error of Mean 5.9 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Test type: Superiority or Other; p = 0.529, Chi-squared; Estimated rate difference = 3.9, 95% CI 2-sided [-8.3 to 16.1], Standard Error of Mean 6.2 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference

3. Primary Outcome: Least Squares Means of Measured Glomerular Filtration Rate (GFR) (Iohexol Serum Clearance in Milliliters Per Minute [mL/Min])
Description: Glomerular filtration rate (GFR): an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using iohexol serum clearance. For determination of iohexol serum clearance, iohexol was administered as an intravenous (IV) bolus over 5 minutes immediately after morning dosing of Tofacitinib or CsA on day of GFR evaluation. Blood samples for iohexol (3 millilitres [mL] each to provide a minimum of 1 mL serum) were collected into appropriately labeled tubes containing no additives at 120, 180, 240, and 300 minutes after the end of the iohexol IV bolus. A normal GFR is greater than (>) 90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR less than (<) 15 mL/min indicated kidney failure.
Time Frame: Month 36
Population: Full analysis set (FAS, which was defined the same as the Safety Analysis Set). The analysis included 1 participant in CsA and 2 in Tofacitinib LI from before protocol Amendment 1. Only subjects at Month 36 with GFR calculations were included.
Measure: Least Squares Mean (Standard Error); unit: mL/min
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 39 | 30 | 13
mL/min | 67.63 (3.38) | 76.86 (3.74) | 75.86 (5.35)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Test type: Superiority or Other; p = 0.0699, Mixed Models Analysis; Mean Difference (Final Values) = 9.23, 60% CI 2-sided [4.97 to 13.49], Standard Error of Mean 5.04 — Tofacitinib LI minus CsA
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Test type: Superiority or Other; p = 0.1958, Mixed Models Analysis; Mean Difference (Final Values) = 8.23, 60% CI 2-sided [2.89 to 13.58], Standard Error of Mean 6.32 — Tofacitinib MI minus CsA

4. Primary Outcome: Percentage of Participants With Progression of Chronic Allograft Lesions at Month 36
Description: Progression of chronic allograft lesions was defined as an increase in the Banff chronicity score (Banff-CS) in biopsy from the implantation (baseline) biopsy in a given participant. Banff-CS was the sum of the Banff scores for the 4 chronic basic lesions (allograft glomerulopathy [cg] + interstitial fibrosis [ci] + tubular atrophy [ct] + vascular intimal thickening [cv]). The Banff-CS ranged from 0-12, higher score indicated greater lesions and Month 36 Banff-CS greater than the implantation biopsy score indicated progression of lesions.
Time Frame: Month 36
Population: FAS. Only participants with Banff CS values at both Day 0 and Month 36 visits were included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 24 | 18 | 8
Percentage of Participants | 87.50 | 77.78 | 87.50

5. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With First Biopsy Proven Acute Rejection (BPAR) by Visit
Description: BPAR was category acute rejection as interpreted by the central blinded pathologist according to the Banff 97 working classification. The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: FAS. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 60 | 54 | 51
Percentage of Participants
  Month 12 | 6.25 [3.70 to 8.80] | 10.00 [6.74 to 13.26] | 5.56 [2.93 to 8.18]
  Month 15 (n=59,54,50) | 7.81 [4.99 to 10.64] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 18 (n=57,54,48) | 9.40 [6.33 to 12.48] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 24 (n=55,53,42) | 9.40 [6.33 to 12.48] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 30 (n=51,37,28) | 9.40 [6.33 to 12.48] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 36 (n=48,28,14) | 11.18 [7.82 to 14.54] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 42 (n=40,28,13) | 13.34 [9.61 to 17.08] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 48 (n=38,28,13) | 13.34 [9.61 to 17.08] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 54 (n=38,27,12) | 13.34 [9.61 to 17.08] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 60 (n=36,23,11) | 13.34 [9.61 to 17.08] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 66 (n=31,20,10) | 13.34 [9.61 to 17.08] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
  Month 72 (n=28,18,10) | 13.34 [9.61 to 17.08] | 10.00 [6.74 to 13.26] | 7.41 [4.41 to 10.41]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.6694, Wald Test; Estimated rate difference = 2.19, 60% CI 2-sided [-2.12 to 6.50], Standard Error of Mean 5.12 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.9340, Wald Test; Estimated rate difference = -0.41, 60% CI 2-sided [-4.52 to 3.71], Standard Error of Mean 4.89 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.9106, Wald Test; Estimated rate difference = 0.60, 60% CI 2-sided [-3.88 to 5.08], Standard Error of Mean 5.32 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.6960, Wald Test; Estimated rate difference = -1.99, 60% CI 2-sided [-6.29 to 2.30], Standard Error of Mean 5.10 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.9106, Wald Test; Estimated rate difference = 0.60, 60% CI 2-sided [-3.88 to 5.08], Standard Error of Mean 5.32 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.6960, Wald Test; Estimated rate difference = -1.99, 60% CI 2-sided [-6.29 to 2.30], Standard Error of Mean 5.10 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.9106, Wald Test; Estimated rate difference = 0.60, 60% CI 2-sided [-3.88 to 5.08], Standard Error of Mean 5.32 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.6960, Wald Test; Estimated rate difference = -1.99, 60% CI 2-sided [-6.29 to 2.30], Standard Error of Mean 5.10 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.8322, Wald Test; Estimated rate difference = -1.18, 60% CI 2-sided [-5.86 to 3.50], Standard Error of Mean 5.56 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.4809, Wald Test; Estimated rate difference = -3.77, 60% CI 2-sided [-8.27 to 0.73], Standard Error of Mean 5.35 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.5704, Wald Test; Estimated rate difference = -3.34, 60% CI 2-sided [-8.31 to 1.62], Standard Error of Mean 5.89 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.2972, Wald Test; Estimated rate difference = -5.94, 60% CI 2-sided [-10.73 to -1.14], Standard Error of Mean 5.70 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.5704, Wald Test; Estimated rate difference = -3.34, 60% CI 2-sided [-8.31 to 1.62], Standard Error of Mean 5.89 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.2972, Wald Test; Estimated rate difference = -5.94, 60% CI 2-sided [-10.73 to -1.14], Standard Error of Mean 5.70 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.5704, Wald Test; Estimated rate difference = -3.34, 60% CI 2-sided [-8.31 to 1.62], Standard Error of Mean 5.89 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.2972, Wald Test; Estimated rate difference = -5.94, 60% CI 2-sided [-10.73 to -1.14], Standard Error of Mean 5.70 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.5704, Wald Test; Estimated rate difference = -3.34, 60% CI 2-sided [-8.31 to 1.62], Standard Error of Mean 5.89 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.2972, Wald Test; Estimated rate difference = -5.94, 60% CI 2-sided [-10.73 to -1.14], Standard Error of Mean 5.70 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.5704, Wald Test; Estimated rate difference = -3.34, 60% CI 2-sided [-8.31 to 1.62], Standard Error of Mean 5.89 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.2972, Wald Test; Estimated rate difference = -5.94, 60% CI 2-sided [-10.73 to -1.14], Standard Error of Mean 5.70 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.5704, Wald Test; Estimated rate difference = -3.34, 60% CI 2-sided [-8.31 to 1.62], Standard Error of Mean 5.89 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.2972, Wald Test; Estimated rate difference = -5.94, 60% CI 2-sided [-10.73 to -1.14], Standard Error of Mean 5.70 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 12; Test type: Superiority or Other; p = 0.4455, Wald Test; Estimated rate difference = 3.75, 60% CI 2-sided [-0.39 to 7.89], Standard Error of Mean 4.91 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 12; Test type: Superiority or Other; p = 0.8730, Wald Test; Estimated rate difference = -0.69, 60% CI 2-sided [-4.35 to 2.96], Standard Error of Mean 4.34 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference

6. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Treated Clinical Acute Rejection by Visit
Description: Treated clinical acute rejection was defined as an acute rejection episode that was diagnosed based on local biopsy readout and received anti-rejection treatment. The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: FAS. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 55 | 56 | 49
Percentage of Participants
  Month 12 | 14.06 [10.41 to 17.72] | 6.67 [3.96 to 9.38] | 9.26 [5.94 to 12.58]
  Month 15 (n=53,56,48) | 17.19 [13.22 to 21.16] | 6.67 [3.96 to 9.38] | 11.11 [7.51 to 14.71]
  Month 18 (n=51,54,46) | 18.75 [14.64 to 22.86] | 10.00 [6.74 to 13.26] | 11.11 [7.51 to 14.71]
  Month 24 (n=49,52,40) | 18.75 [14.64 to 22.86] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 30 (n=46,37,27) | 20.48 [16.21 to 24.75] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 36 (n=42,29,14) | 23.94 [19.38 to 28.49] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 42 (n=36,29,13) | 27.56 [22.74 to 32.38] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 48 (n=34,29,13) | 27.56 [22.74 to 32.38] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 54 (n=33,28,12) | 29.69 [24.69 to 34.69] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 60 (n=30,24,11) | 29.69 [24.69 to 34.69] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 66 (n=25,21,9) | 29.69 [24.69 to 34.69] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
  Month 72 (n=22,18,9) | 29.69 [24.69 to 34.69] | 11.67 [8.18 to 15.15] | 11.11 [7.51 to 14.71]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.0654, Wald Test; Estimated rate difference = -10.52, 60% CI 2-sided [-15.33 to -5.71], Standard Error of Mean 5.71 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.3398, Wald Test; Estimated rate difference = -6.08, 60% CI 2-sided [-11.43 to -0.72], Standard Error of Mean 6.37 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.1601, Wald Test; Estimated rate difference = -8.75, 60% CI 2-sided [-13.99 to -3.51], Standard Error of Mean 6.23 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.2390, Wald Test; Estimated rate difference = -7.64, 60% CI 2-sided [-13.10 to -2.18], Standard Error of Mean 6.49 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.2685, Wald Test; Estimated rate difference = -7.08, 60% CI 2-sided [-12.47 to -1.70], Standard Error of Mean 6.40 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.2390, Wald Test; Estimated rate difference = -7.64, 60% CI 2-sided [-13.10 to -2.18], Standard Error of Mean 6.49 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.1785, Wald Test; Estimated rate difference = -8.81, 60% CI 2-sided [-14.32 to -3.30], Standard Error of Mean 6.55 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.1580, Wald Test; Estimated rate difference = -9.37, 60% CI 2-sided [-14.95 to -3.78], Standard Error of Mean 6.63 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.0718, Wald Test; Estimated rate difference = -12.27, 60% CI 2-sided [-18.00 to -6.53], Standard Error of Mean 6.81 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.0629, Wald Test; Estimated rate difference = -12.83, 60% CI 2-sided [-18.63 to -7.02], Standard Error of Mean 6.90 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0246, Wald Test; Estimated rate differences = -15.89, 60% CI 2-sided [-21.84 to -9.94], Standard Error of Mean 7.07 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.0214, Wald Test; Estimated rate difference = -16.45, 60% CI 2-sided [-22.46 to -10.43], Standard Error of Mean 7.15 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0246, Wald Test; Estimated rate difference = -15.89, 60% CI 2-sided [-21.84 to -9.94], Standard Error of Mean 7.07 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.0214, Wald Test; Estimated rate difference = -16.45, 60% CI 2-sided [-22.46 to -10.43], Standard Error of Mean 7.15 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0128, Wald Test; Estimated rate difference = -18.02, 60% CI 2-sided [-24.12 to -11.93], Standard Error of Mean 7.24 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.0111, Wald Test; Estimated rate difference = -18.58, 60% CI 2-sided [-24.74 to -12.42], Standard Error of Mean 7.32 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0128, Wald Test; Estimated rate difference = -18.02, 60% CI 2-sided [-24.12 to -11.93], Standard Error of Mean 7.24 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.0111, Wald Test; Estimated rate difference = -18.58, 60% CI 2-sided [-24.74 to -12.42], Standard Error of Mean 7.32 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0128, Wald Test; Estimated rate difference = -18.02, 60% CI 2-sided [-24.12 to -11.93], Standard Error of Mean 7.24 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.0111, Wald Test; Estimated rate difference = -18.58, 60% CI 2-sided [-24.74 to -12.42], Standard Error of Mean 7.32 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0128, Wald Test; Estimated rate difference = -18.02, 60% CI 2-sided [-24.12 to -11.93], Standard Error of Mean 7.24 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.0111, Wald Test; Estimated rate difference = -18.58, 60% CI 2-sided [-24.74 to -12.42], Standard Error of Mean 7.32 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 12; Test type: Superiority or Other; p = 0.1715, Wald Test; Estimated rate difference = -7.40, 60% CI 2-sided [-11.95 to -2.84], Standard Error of Mean 5.41 — Tofacitinib LI minus CsA Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 12; Test type: Superiority or Other; p = 0.4131, Wald Test; Estimated rate difference = -4.80, 60% CI 2-sided [-9.74 to 0.14], Standard Error of Mean 5.87 — Tofacitinib MI minus CsA Standard error of the mean refers to standard error of the estimated rate difference

7. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Efficacy Failure by Visit
Description: Efficacy failure was the first occurrence of BPAR diagnosed by the central pathologist or graft loss including participant death. BPAR (category acute rejection) was interpreted by the central blinded pathologist according to the Banff 97 working classification. The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: FAS. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 60 | 54 | 51
Percentage of Participants
  Month 12 | 6.25 [3.70 to 8.80] | 10.00 [6.74 to 13.26] | 5.56 [2.93 to 8.18]
  Month 15 (n=58,54,49) | 7.81 [4.99 to 10.64] | 10.00 [6.74 to 13.26] | 9.26 [5.94 to 12.58]
  Month 18 (n=56,54,49) | 10.99 [7.69 to 14.29] | 10.00 [6.74 to 13.26] | 9.26 [5.94 to 12.58]
  Month 24 (n=54,54,46) | 10.99 [7.69 to 14.29] | 10.00 [6.74 to 13.26] | 14.81 [10.75 to 18.88]
  Month 30 (n=53,52,46) | 12.64 [9.12 to 16.16] | 10.00 [6.74 to 13.26] | 14.81 [10.75 to 18.88]
  Month 36 (n=51,48,42) | 15.94 [12.04 to 19.83] | 15.19 [11.26 to 19.12] | 16.71 [12.43 to 20.99]
  Month 42 (n=44,47,41) | 19.59 [15.30 to 23.88] | 15.19 [11.26 to 19.12] | 18.69 [14.20 to 23.18]
  Month 48 (n=43,44,38) | 21.42 [16.96 to 25.88] | 18.84 [14.52 to 23.16] | 18.69 [14.20 to 23.18]
  Month 54 (n=41,44,36) | 23.25 [18.63 to 27.86] | 18.84 [14.52 to 23.16] | 18.69 [14.20 to 23.18]
  Month 60 (n=41,44,35) | 23.25 [18.63 to 27.86] | 18.84 [14.52 to 23.16] | 20.95 [16.20 to 25.70]
  Month 66 (n=39,42,29) | 23.25 [18.63 to 27.86] | 18.84 [14.52 to 23.16] | 20.95 [16.20 to 25.70]
  Month 72 (n=35,28,19) | 23.25 [18.63 to 27.86] | 22.81 [18.10 to 27.51] | 20.95 [16.20 to 25.70]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.6694, Wald Test; Estimated rate difference = 2.19, 60% CI 2-sided [-2.12 to 6.50], Standard Error of Mean 5.12 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.7799, Wald Test; Estimated rate difference = 1.45, 60% CI 2-sided [-2.91 to 5.80], Standard Error of Mean 5.18 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.8572, Wald Test; Estimated rate difference = -0.99, 60% CI 2-sided [-5.63 to 3.65], Standard Error of Mean 5.51 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.7555, Wald Test; Estimated rate difference = -1.73, 60% CI 2-sided [-6.41 to 2.95], Standard Error of Mean 5.56 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.8572, Wald Test; Estimated rate difference = -0.99, 60% CI 2-sided [-5.63 to 3.65], Standard Error of Mean 5.51 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.5390, Wald Test; Estimated rate difference = 3.82, 60% CI 2-sided [-1.41 to 9.06], Standard Error of Mean 6.22 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.6432, Wald Test; Estimated rate difference = -2.64, 60% CI 2-sided [-7.44 to 2.16], Standard Error of Mean 5.70 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.7336, Wald Test; Estimated rate difference = 2.18, 60% CI 2-sided [-3.20 to 7.55], Standard Error of Mean 6.39 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.9099, Wald Test; Estimated rate difference = -0.74, 60% CI 2-sided [-6.28 to 4.79], Standard Error of Mean 6.57 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.9106, Wald Test; Estimated rate difference = 0.77, 60% CI 2-sided [-5.01 to 6.56], Standard Error of Mean 6.87 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.5244, Wald Test; Estimated rate difference = -4.40, 60% CI 2-sided [-10.22 to 1.42], Standard Error of Mean 6.91 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.9029, Wald Test; Estimated rate difference = -0.90, 60% CI 2-sided [-7.11 to 5.31], Standard Error of Mean 7.38 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.7267, Wald Test; Estimated rate difference = -2.58, 60% CI 2-sided [-8.78 to 3.63], Standard Error of Mean 7.38 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.7168, Wald Test; Estimated rate difference = -2.73, 60% CI 2-sided [-9.06 to 3.60], Standard Error of Mean 7.52 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.5574, Wald Test; Estimated rate difference = -4.40, 60% CI 2-sided [-10.72 to 1.91], Standard Error of Mean 7.51 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.5515, Wald Test; Estimated rate difference = -4.56, 60% CI 2-sided [-10.99 to 1.88], Standard Error of Mean 7.65 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.5574, Wald Test; Estimated rate difference = -4.40, 60% CI 2-sided [-10.72 to 1.91], Standard Error of Mean 7.51 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.7704, Wald Test; Estimated rate difference = -2.30, 60% CI 2-sided [-8.92 to 4.33], Standard Error of Mean 7.87 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.5574, Wald Test; Estimated rate difference = -4.40, 60% CI 2-sided [-10.72 to 1.91], Standard Error of Mean 7.51 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.7704, Wald Test; Estimated rate difference = -2.30, 60% CI 2-sided [-8.92 to 4.33], Standard Error of Mean 7.87 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.9551, Wald Test; Estimated rate difference = -0.44, 60% CI 2-sided [-7.03 to 6.15], Standard Error of Mean 7.83 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.7704, Wald Test; Estimated rate difference = -2.30, 60% CI 2-sided [-8.92 to 4.33], Standard Error of Mean 7.87 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 12; Test type: Superiority or Other; p = 0.4455, Wald Test; Mean Difference (Final Values) = 3.75, 60% CI 2-sided [-0.39 to 7.89], Standard Error of Mean 4.91
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 12; Test type: Superiority or Other; p = 0.8730, Wald Test; Estimated rate difference = -0.69, 60% CI 2-sided [-4.35 to 2.96], Standard Error of Mean 4.34 — Standard error of the mean refers to standard error of the estimated rate difference

8. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Combined Banff Rejection by Visit
Description: Banff 97: standard classification for scoring and classifying rejection of kidney transplant biopsies in 6 diagnostic categories: normal, antibody-mediated rejection, borderline changes: 'suspicious' for acute cellular rejection, acute/active cellular rejection, chronic/sclerosing allograft nephropathy, and other. Combined Banff rejection was calculated from categories of antibody-mediated rejection (Category 2) plus borderline changes (Category 3) plus acute rejection (Category 4), as interpreted by the central pathologist. The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: FAS. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 54 | 52 | 48
Percentage of Participants
  Month 12 | 15.63 [11.81 to 19.44] | 13.33 [9.64 to 17.03] | 11.11 [7.51 to 14.71]
  Month 15 (n=51,52,45) | 20.31 [16.08 to 24.55] | 13.33 [9.64 to 17.03] | 16.67 [12.40 to 20.93]
  Month 18 (n=49,52,43) | 21.91 [17.55 to 26.26] | 13.33 [9.64 to 17.03] | 16.67 [12.40 to 20.93]
  Month 24 (n=46,50,37) | 23.57 [19.09 to 28.05] | 15.00 [11.12 to 18.88] | 18.60 [14.13 to 23.07]
  Month 30 (n=44,37,23) | 23.57 [19.09 to 28.05] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 36 (n=41,28,12) | 25.30 [20.69 to 29.92] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 42 (n=34,28,11) | 27.44 [22.62 to 32.26] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 48 (n=33,28,11) | 27.44 [22.62 to 32.26] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 54 (n=33,27,10) | 27.44 [22.62 to 32.26] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 60 (n=31,23,9) | 27.44 [22.62 to 32.26] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 66 (n=26,20,9) | 27.44 [22.62 to 32.26] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
  Month 72 (n=24,18,9) | 27.44 [22.62 to 32.26] | 15.00 [11.12 to 18.88] | 21.41 [16.51 to 26.31]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.2957, Wald Test; Estimated rate difference = -6.98, 60% CI 2-sided [-12.60 to -1.36], Standard Error of Mean 6.67 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.6097, Wald Test; Estimated rate difference = -3.65, 60% CI 2-sided [-9.66 to 2.37], Standard Error of Mean 7.14 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.2064, Wald Test; Estimated rate difference = -8.57, 60% CI 2-sided [-14.28 to -2.86], Standard Error of Mean 6.79 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.4696, Wald Test; Estimated rate difference = -5.24, 60% CI 2-sided [-11.34 to 0.86], Standard Error of Mean 7.25 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.2238, Wald Test; Estimated rate difference = -8.57, 60% CI 2-sided [-14.50 to -2.64], Standard Error of Mean 7.04 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.5093, Wald Test; Estimated rate difference = -4.96, 60% CI 2-sided [-11.29 to 1.37], Standard Error of Mean 7.52 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.2238, Wald Test; Estimated rate difference = -8.57, 60% CI 2-sided [-14.50 to -2.64], Standard Error of Mean 7.04 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.7846, Wald Test; Estimated rate difference = -2.16, 60% CI 2-sided [-8.80 to 4.48], Standard Error of Mean 7.89 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.1501, Wald Test; Estimated rate difference = -10.30, 60% CI 2-sided [-16.33 to -4.28], Standard Error of Mean 7.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.6263, Wald Test; Estimated rate difference = -3.89, 60% CI 2-sided [-10.62 to 2.84], Standard Error of Mean 8.00 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0905, Wald Test; Estimated rate difference = -12.44, 60% CI 2-sided [-18.62 to -6.25], Standard Error of Mean 7.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.4604, Wald Test; Estimated rate difference = -6.03, 60% CI 2-sided [-12.90 to 0.84], Standard Error of Mean 8.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0905, Wald Test; Estimated rate difference = -12.44, 60% CI 2-sided [-18.62 to -6.25], Standard Error of Mean 7.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.4604, Wald Test; Estimated rate difference = -6.03, 60% CI 2-sided [-12.90 to 0.84], Standard Error of Mean 8.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0905, Wald Test; Estimated rate difference = -12.44, 60% CI 2-sided [-18.62 to -6.25], Standard Error of Mean 7.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.4604, Wald Test; Estimated rate difference = -6.03, 60% CI 2-sided [-12.90 to 0.84], Standard Error of Mean 8.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0905, Wald Test; Estimated rate difference = -12.44, 60% CI 2-sided [-18.62 to -6.25], Standard Error of Mean 7.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.4604, Wald Test; Estimated rate difference = -6.03, 60% CI 2-sided [-12.90 to 0.84], Standard Error of Mean 8.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0905, Wald Test; Estimated rate difference = -12.44, 60% CI 2-sided [-18.62 to -6.25], Standard Error of Mean 7.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.4604, Wald Test; Estimated rate difference = -6.03, 60% CI 2-sided [-12.90 to 0.84], Standard Error of Mean 8.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0905, Wald Test; Estimated rate difference = -12.44, 60% CI 2-sided [-18.62 to -6.25], Standard Error of Mean 7.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.4604, Wald Test; Estimated rate difference = -6.03, 60% CI 2-sided [-12.90 to 0.84], Standard Error of Mean 8.16 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 12; Test type: Superiority or Other; p = 0.7166, Wald Test; Estimated rate difference = -2.29, 60% CI 2-sided [-7.61 to 3.02], Standard Error of Mean 6.31 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 12; Test type: Superiority or Other; p = 0.4692, Wald Test; Estimated rate difference = -4.51, 60% CI 2-sided [-9.76 to 0.73], Standard Error of Mean 6.24 — Standard error of the mean refers to standard error of the estimated rate difference

9. Secondary Outcome: Kaplan-Meier Analysis of Percent of Participants With Graft Survival With Death Censored by Visit
Description: Graft loss was defined as graft nephrectomy, subject death, retransplantation, or return to dialysis for at least 6 consecutive weeks. The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits. Included data up to 2 months postdose in the clinical Follow-up visit.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: FAS. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 64 | 60 | 54
Percentage of participants
  Month 12 | 100.00 [99.58 to 100.00] | 100.00 [98.48 to 100.00] | 100.00 [98.32 to 100.00]
  Month 15 | 100.00 [95.58 to 100.00] | 100.00 [98.48 to 100.00] | 100.00 [98.32 to 100.00]
  Month 18 (n=62,59,51) | 100.00 [98.53 to 100.00] | 100.00 [98.46 to 100.00] | 100.00 [98.22 to 100.00]
  Month 24 (n=59,58,45) | 100.00 [98.46 to 100.00] | 100.00 [98.43 to 100.00] | 100.00 [97.98 to 100.00]
  Month 30 (n=55,42,31) | 98.31 [96.89 to 99.72] | 100.00 [97.84 to 100.00] | 100.00 [97.09 to 100.00]
  Month 36 (n=53,32,16) | 96.48 [94.43 to 98.54] | 100.00 [97.18 to 100.00] | 100.00 [94.43 to 100.00]
  Month 42 (n=46,32,15) | 96.48 [94.43 to 98.54] | 100.00 [97.18 to 100.00] | 100.00 [94.07 to 100.00]
  Month 48 (n=44,32,15) | 96.48 [94.43 to 98.54] | 100.00 [97.18 to 100.00] | 100.00 [94.07 to 100.00]
  Month 54 (n=43,31,14) | 96.48 [94.43 to 98.54] | 100.00 [97.09 to 100.00] | 100.00 [93.66 to 100.00]
  Month 60 (n=40,26,13) | 96.48 [94.43 to 98.54] | 100.00 [96.54 to 100.00] | 100.00 [93.19 to 100.00]
  Month 66 (n=35,23,11) | 96.48 [94.43 to 98.54] | 100.00 [96.09 to 100.00] | 100.00 [92.01 to 100.00]
  Month 72 (n=31,20,11) | 96.48 [94.43 to 98.54] | 100.00 [95.52 to 100.00] | 100.00 [92.01 to 100.00]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.3132, Wald Test; Estimated rate difference = 1.69, 60% CI 2-sided [0.28 to 3.11], Standard Error of Mean 1.68 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.3132, Wald Test; Estimated rate difference = 1.69, 60% CI 2-sided [0.28 to 3.11], Standard Error of Mean 1.68 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.1503, Wald Test; Estimated rate difference = 3.52, 60% CI 2-sided [1.46 to 5.57], Standard Error of Mean 2.44 — Standard error of the mean refers to standard error of the estimated rate difference

10. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants Surviving by Visit
Description: The 'Number' and 'Other Confidence Interval Level' columns represent cumulative proportions and 60% confidence intervals (CIs) as estimated from the fitted Kaplan-Meier curves for each treatment at scheduled visits. Included data up to 2 months postdose in the clinical Follow-up visit.
Time Frame: Months 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: FAS. n is the number of participants remaining at risk at each visit.
Measure: Number (60% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 64 | 60 | 54
Percentage of Participants
  Month 12 | 100.00 [98.58 to 100.00] | 100.00 [98.48 to 100.00] | 100.00 [98.32 to 100.00]
  Month 15 (n=64,60,53) | 100.00 [98.58 to 100.00] | 100.00 [98.48 to 100.00] | 98.15 [96.60 to 99.69]
  Month 18 (n=61,59,51) | 98.41 [97.09 to 99.74] | 100.00 [98.46 to 100.00] | 98.15 [96.60 to 99.69]
  Month 24 (n=59,58,44) | 98.41 [97.09 to 99.74] | 100.00 [98.43 to 100.00] | 94.22 [91.49 to 96.95]
  Month 30 (n=55,42,31) | 98.41 [97.09 to 99.74] | 100.00 [97.84 to 100.00] | 94.22 [91.49 to 96.95]
  Month 36 (n=53,32,16) | 98.41 [97.09 to 99.74] | 100.00 [97.18 to 100.00] | 90.97 [87.21 to 94.73]
  Month 42 (n=45,32,15) | 96.27 [94.07 to 98.48] | 100.00 [97.18 to 100.00] | 90.97 [87.21 to 94.73]
  Month 48 (n=44,32,15) | 96.27 [94.07 to 98.48] | 100.00 [97.18 to 100.00] | 90.97 [87.21 to 94.73]
  Month 54 (n=43,31,14) | 94.09 [91.27 to 96.90] | 100.00 [97.09 to 100.00] | 90.97 [87.21 to 94.73]
  Month 60 (n=40,26,13) | 94.09 [91.27 to 96.90] | 100.00 [96.54 to 100.00] | 90.97 [87.21 to 94.73]
  Month 66 (n=35,23,11) | 94.09 [91.27 to 96.90] | 100.00 [96.09 to 100.00] | 90.97 [87.21 to 94.73]
  Month 72 (n=31,20,11) | 94.09 [91.27 to 96.90] | 100.00 [95.52 to 100.00] | 90.97 [87.21 to 94.73]
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.3128, Wald Test; Estimated rate difference = -1.85, 60% CI 2-sided [-3.40 to -0.31], Standard Error of Mean 1.83 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.3134, Wald Test; Estimated rate difference = 1.59, 60% CI 2-sided [0.26 to 2.91], Standard Error of Mean 1.57 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.9129, Wald Test; Estimated rate difference = -0.26, 60% CI 2-sided [-2.30 to 1.77], Standard Error of Mean 2.42 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.3134, Wald Test; Estimated rate difference = 1.59, 60% CI 2-sided [0.26 to 2.91], Standard Error of Mean 1.57 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.2447, Wald Test; Estimated rate difference = -4.19, 60% CI 2-sided [-7.23 to -1.16], Standard Error of Mean 3.61 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.3134, Wald Test; Estimated rate difference = 1.59, 60% CI 2-sided [0.26 to 2.91], Standard Error of Mean 1.57 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.2447, Wald Test; Estimated rate difference = -4.19, 60% CI 2-sided [-7.23 to -1.16], Standard Error of Mean 3.61 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.3134, Wald Test; Estimated rate difference = 1.59, 60% CI 2-sided [0.26 to 2.91], Standard Error of Mean 1.57 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.1164, Wald Test; Estimated rate difference = -7.44, 60% CI 2-sided [-11.43 to -3.45], Standard Error of Mean 4.74 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.1545, Wald Test; Estimated rate difference = 3.73, 60% CI 2-sided [1.52 to 5.93], Standard Error of Mean 2.62 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.3061, Wald Test; Estimated rate difference = -5.30, 60% CI 2-sided [-9.66 to -0.94], Standard Error of Mean 5.18 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.1545, Wald Test; Estimated rate difference = 3.73, 60% CI 2-sided [1.52 to 5.93], Standard Error of Mean 2.62 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.3061, Wald Test; Estimated rate difference = -5.30, 60% CI 2-sided [-9.66 to -0.94], Standard Error of Mean 5.18 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0774, Wald Test; Estimated rate difference = 5.91, 60% CI 2-sided [3.10 to 8.73], Standard Error of Mean 3.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.5772, Wald Test; Estimated rate difference = -3.12, 60% CI 2-sided [-7.82 to 1.59], Standard Error of Mean 5.59 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0774, Wald Test; Estimated rate difference = 5.91, 60% CI 2-sided [3.10 to 8.73], Standard Error of Mean 3.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.5772, Wald Test; Estimated rate difference = -3.12, 60% CI 2-sided [-7.82 to 1.59], Standard Error of Mean 5.59 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0774, Wald Test; Estimated rate difference = 5.91, 60% CI 2-sided [3.10 to 8.73], Standard Error of Mean 3.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.5772, Wald Test; Estimated rate difference = -3.12, 60% CI 2-sided [-7.82 to 1.59], Standard Error of Mean 5.59 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0774, Wald Test; Estimated rate difference = 5.91, 60% CI 2-sided [3.10 to 8.73], Standard Error of Mean 3.35 — Standard error of the mean refers to standard error of the estimated rate difference
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.5772, Wald Test; Estimated rate difference = -3.12, 60% CI 2-sided [-7.82 to 1.59], Standard Error of Mean 5.59 — Standard error of the mean refers to standard error of the estimated rate difference

11. Secondary Outcome: Percentage of Participants Discontinuing From the Study
Description: Discontinuations were due to any reason including those occurring as a result of protocol Amendments 3 and 4.
Time Frame: Months 12 through 72.
Population: Safety Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 64 | 60 | 54
Percentage of Participants | 43.8 | 75.0 | 85.2

12. Secondary Outcome: Least Squares Means of Total Serum Cholesterol Levels (Milligrams Per Deciliter [mg/dL]) by Visit
Description: Model contained treatment, visit and treatment by visit interaction as fixed effects and Baseline (predose in Study A3921030) as a covariate. A first-order autoregressive variance-covariance structure was used.
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 49
mg/dL
  Month 15 | 199.14 (5.71) | 213.49 (5.81) | 196.27 (6.29)
  Month 18 | 200.51 (5.75) | 212.67 (5.82) | 193.50 (6.34)
  Month 24 (n=58,54,40) | 198.78 (5.82) | 212.30 (5.98) | 185.57 (6.80)
  Month 30 (n=52,37,26) | 193.99 (6.05) | 211.59 (6.84) | 202.73 (8.08)
  Month 36 (n=51,32,15) | 198.62 (6.17) | 211.14 (7.51) | 192.97 (10.37)
  Month 42 (n=44,31,15) | 200.36 (6.52) | 220.29 (7.83) | 208.77 (11.13)
  Month 48 (n=42,30,14) | 196.56 (6.74) | 228.83 (7.98) | 188.83 (11.66)
  Month 54 (n=41,31,13) | 193.66 (6.87) | 222.86 (7.98) | 183.17 (12.06)
  Month 60 (n=37,23,12) | 190.10 (7.17) | 220.47 (8.85) | 184.14 (12.53)
  Month 66 (n=34,20,11) | 191.00 (7.47) | 218.77 (9.47) | 189.15 (13.14)
  Month 72 (n=31,17,11) | 188.74 (7.82) | 209.12 (10.26) | 182.60 (13.36)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.0786, Mixed Models Analysis; Mean Difference (Final Values) = 14.35, 60% CI 2-sided [7.49 to 21.22], Standard Error of Mean 8.15
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.7360, Mixed Models Analysis; Mean Difference (Final Values) = -2.87, 60% CI 2-sided [-10.03 to 4.29], Standard Error of Mean 8.50
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.1377, Mixed Models Analysis; Mean Difference (Final Values) = 12.16, 60% CI 2-sided [5.27 to 19.05], Standard Error of Mean 8.19
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.4131, Mixed Models Analysis; Mean Difference (Final Values) = -7.01, 60% CI 2-sided [-14.21 to 0.20], Standard Error of Mean 8.56
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.1057, Mixed Models Analysis; Mean Difference (Final Values) = 13.52, 60% CI 2-sided [6.49 to 20.55], Standard Error of Mean 8.35
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.1402, Mixed Models Analysis; Mean Difference (Final Values) = -13.21, 60% CI 2-sided [-20.75 to -5.68], Standard Error of Mean 8.95
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.0542, Mixed Models Analysis; Mean Difference (Final Values) = 17.60, 60% CI 2-sided [9.91 to 25.29], Standard Error of Mean 9.13
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.3866, Mixed Models Analysis; Mean Difference (Final Values) = 8.74, 60% CI 2-sided [0.24 to 17.24], Standard Error of Mean 10.09
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.1981, Mixed Models Analysis; Mean Difference (Final Values) = 12.52, 60% CI 2-sided [4.33 to 20.71], Standard Error of Mean 9.72
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.6397, Mixed Models Analysis; Mean Difference (Final Values) = -5.65, 60% CI 2-sided [-15.81 to 4.51], Standard Error of Mean 12.07
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0508, Mixed Models Analysis; Mean Difference (Final Values) = 19.93, 60% CI 2-sided [11.35 to 28.51], Standard Error of Mean 10.19
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.5143, Mixed Models Analysis; Mean Difference (Final Values) = 8.42, 60% CI 2-sided [-2.45 to 19.28], Standard Error of Mean 12.90
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; Mean Difference (Final Values) = 32.26, 60% CI 2-sided [23.46 to 41.06], Standard Error of Mean 10.45
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.5661, Mixed Models Analysis; Mean Difference (Final Values) = -7.73, 60% CI 2-sided [-19.07 to 3.61], Standard Error of Mean 13.47
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0057, Mixed Models Analysis; Mean Difference (Final Values) = 29.20, 60% CI 2-sided [20.33 to 38.08], Standard Error of Mean 10.54
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.4504, Mixed Models Analysis; Mean Difference (Final Values) = -10.49, 60% CI 2-sided [-22.18 to 1.21], Standard Error of Mean 13.89
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0078, Mixed Models Analysis; Mean Difference (Final Values) = 30.37, 60% CI 2-sided [20.78 to 39.96], Standard Error of Mean 11.39
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.6802, Mixed Models Analysis; Mean Difference (Final Values) = -5.95, 60% CI 2-sided [-18.11 to 6.20], Standard Error of Mean 14.44
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0216, Mixed Models Analysis; Mean Difference (Final Values) = 27.78, 60% CI 2-sided [17.61 to 37.95], Standard Error of Mean 12.08
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.9026, Mixed Models Analysis; Mean Difference (Final Values) = -1.85, 60% CI 2-sided [-14.58 to 10.88], Standard Error of Mean 15.12
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.1146, Mixed Models Analysis; Mean Difference (Final Values) = 20.38, 60% CI 2-sided [9.51 to 31.24], Standard Error of Mean 12.91
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.6918, Mixed Models Analysis; Mean Difference (Final Values) = -6.14, 60% CI 2-sided [-19.18 to 6.90], Standard Error of Mean 15.48

13. Secondary Outcome: Least Squares Means of Total Serum Low Density Lipoprotein (LDL) Cholesterol Levels (mg/dL) by Visit
Description: as for outcome 12
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 56 | 54 | 49
mg/dL
  Month 15 (n=54,54,48) | 113.09 (4.60) | 119.71 (4.68) | 108.72 (4.94)
  Month 18 | 112.82 (4.58) | 119.36 (4.69) | 109.87 (4.94)
  Month 24 (n=55,49,40) | 111.14 (4.64) | 119.15 (4.83) | 104.63 (5.29)
  Month 30 (n=49,36,25) | 106.79 (4.84) | 125.24 (5.43) | 112.44 (6.36)
  Month 36 (n=47,31,15) | 112.81 (4.97) | 123.27 (5.95) | 109.54 (8.10)
  Month 42 (n=42,27,15) | 110.98 (5.21) | 122.51 (6.39) | 121.74 (8.67)
  Month 48 (n=41,27,14) | 109.03 (5.35) | 127.65 (6.48) | 105.59 (9.08)
  Month 54 (n=40,28,13) | 107.21 (5.44) | 128.39 (6.45) | 96.60 (9.39)
  Month 60 (n=36,21,12) | 105.37 (5.66) | 123.71 (7.18) | 97.79 (9.75)
  Month 66 (n=32,19,11) | 104.31 (5.95) | 123.74 (7.64) | 102.44 (10.23)
  Month 72 (n=30,16,11) | 109.18 (6.19) | 116.17 (8.27) | 96.11 (10.40)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.3139, Mixed Models Analysis; Mean Difference (Final Values) = 6.62, 60% CI 2-sided [1.09 to 12.14], Standard Error of Mean 6.57
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.5176, Mixed Models Analysis; Mean Difference (Final Values) = -4.37, 60% CI 2-sided [-10.06 to 1.31], Standard Error of Mean 6.75
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.3191, Mixed Models Analysis; Mean Difference (Final Values) = 6.54, 60% CI 2-sided [1.02 to 12.06], Standard Error of Mean 6.56
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.6608, Mixed Models Analysis; Mean Difference (Final Values) = -2.95, 60% CI 2-sided [-8.62 to 2.71], Standard Error of Mean 6.73
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.2319, Mixed Models Analysis; Mean Difference (Final Values) = 8.02, 60% CI 2-sided [2.37 to 13.66], Standard Error of Mean 6.70
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.3554, Mixed Models Analysis; Mean Difference (Final Values) = -6.50, 60% CI 2-sided [-12.43 to -0.58], Standard Error of Mean 7.04
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.0113, Mixed Models Analysis; Mean Difference (Final Values) = 18.45, 60% CI 2-sided [12.33 to 24.57], Standard Error of Mean 7.27
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.4790, Mixed Models Analysis; Mean Difference (Final Values) = 5.66, 60% CI 2-sided [-1.07 to 12.39], Standard Error of Mean 7.99
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.1776, Mixed Models Analysis; Mean Difference (Final Values) = 10.46, 60% CI 2-sided [3.93 to 16.99], Standard Error of Mean 7.75
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.7307, Mixed Models Analysis; Mean Difference (Final Values) = -3.27, 60% CI 2-sided [-11.27 to 4.73], Standard Error of Mean 9.50
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.1625, Mixed Models Analysis; Mean Difference (Final Values) = 11.53, 60% CI 2-sided [4.59 to 18.48], Standard Error of Mean 8.25
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.2876, Mixed Models Analysis; Mean Difference (Final Values) = 10.77, 60% CI 2-sided [2.25 to 19.29], Standard Error of Mean 10.12
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0270, Mixed Models Analysis; Mean Difference (Final Values) = 18.62, 60% CI 2-sided [11.54 to 25.70], Standard Error of Mean 8.41
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.7444, Mixed Models Analysis; Mean Difference (Final Values) = -3.44, 60% CI 2-sided [-12.31 to 5.44], Standard Error of Mean 10.54
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0122, Mixed Models Analysis; Mean Difference (Final Values) = 21.18, 60% CI 2-sided [14.08 to 28.29], Standard Error of Mean 8.44
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.3288, Mixed Models Analysis; Mean Difference (Final Values) = -10.61, 60% CI 2-sided [-19.75 to -1.47], Standard Error of Mean 10.86
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0453, Mixed Models Analysis; Mean Difference (Final Values) = 18.34, 60% CI 2-sided [10.63 to 26.05], Standard Error of Mean 9.15
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.5016, Mixed Models Analysis; Mean Difference (Final Values) = -7.59, 60% CI 2-sided [-17.09 to 1.91], Standard Error of Mean 11.28
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0453, Mixed Models Analysis; Mean Difference (Final Values) = 19.43, 60% CI 2-sided [11.27 to 27.59], Standard Error of Mean 9.69
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.8747, Mixed Models Analysis; Mean Difference (Final Values) = -1.87, 60% CI 2-sided [-11.83 to 8.10], Standard Error of Mean 11.84
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.4997, Mixed Models Analysis; Mean Difference (Final Values) = 6.98, 60% CI 2-sided [-1.72 to 15.69], Standard Error of Mean 10.34
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.2804, Mixed Models Analysis; Mean Difference (Final Values) = -13.07, 60% CI 2-sided [-23.26 to -2.88], Standard Error of Mean 12.10

14. Secondary Outcome: Least Squares Means of Total Serum High Density Lipoprotein (HDL) Cholesterol Levels (mg/dL) by Visit
Description: as for outcome 12
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 49
mg/dL
  Month 15 | 49.88 (1.75) | 59.67 (1.79) | 55.20 (1.93)
  Month 18 | 50.47 (1.77) | 59.87 (1.79) | 55.78 (1.95)
  Month 24 (n=58,54,40) | 51.47 (1.79) | 59.84 (1.84) | 53.52 (2.08)
  Month 30 (n=52,37,26) | 49.55 (1.85) | 60.45 (2.10) | 53.84 (2.47)
  Month 36 (n=51,32,15) | 50.46 (1.89) | 59.92 (2.30) | 54.59 (3.17)
  Month 42 (n=44,31,15) | 53.24 (2.00) | 59.32 (2.40) | 58.59 (3.41)
  Month 48 (n=42,30,14) | 54.59 (2.07) | 61.67 (2.45) | 53.55 (3.57)
  Month 54 (n=41,31,13) | 54.55 (2.11) | 60.18 (2.45) | 52.38 (3.70)
  Month 60 (n=37,23,12) | 54.72 (2.20) | 60.20 (2.71) | 58.98 (3.84)
  Month 66 (n=34,20,11) | 54.69 (2.29) | 62.12 (2.90) | 56.08 (4.03)
  Month 72 (31,17,11) | 52.80 (2.40) | 58.80 (3.14) | 54.93 (4.10)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 9.79, 60% CI 2-sided [7.68 to 11.90], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.0418, Mixed Models Analysis; Mean Difference (Final Values) = 5.32, 60% CI 2-sided [3.12 to 7.52], Standard Error of Mean 2.61
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 9.40, 60% CI 2-sided [7.28 to 11.51], Standard Error of Mean 2.51
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.0437, Mixed Models Analysis; Mean Difference (Final Values) = 5.30, 60% CI 2-sided [3.09 to 7.51], Standard Error of Mean 2.63
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = 8.37, 60% CI 2-sided [6.21 to 10.53], Standard Error of Mean 2.56
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.4565, Mixed Models Analysis; Mean Difference (Final Values) = 2.04, 60% CI 2-sided [-0.27 to 4.36], Standard Error of Mean 2.75
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 10.90, 60% CI 2-sided [8.54 to 13.26], Standard Error of Mean 2.80
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.1654, Mixed Models Analysis; Mean Difference (Final Values) = 4.29, 60% CI 2-sided [1.69 to 6.89], Standard Error of Mean 3.09
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 9.45, 60% CI 2-sided [6.95 to 11.96], Standard Error of Mean 2.98
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.2636, Mixed Models Analysis; Mean Difference (Final Values) = 4.13, 60% CI 2-sided [1.02 to 7.23], Standard Error of Mean 3.69
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0520, Mixed Models Analysis; Mean Difference (Final Values) = 6.08, 60% CI 2-sided [3.45 to 8.71], Standard Error of Mean 3.12
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.1760, Mixed Models Analysis; Mean Difference (Final Values) = 5.35, 60% CI 2-sided [2.02 to 8.67], Standard Error of Mean 3.95
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0274, Mixed Models Analysis; Mean Difference (Final Values) = 7.08, 60% CI 2-sided [4.38 to 9.77], Standard Error of Mean 3.20
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.8018, Mixed Models Analysis; Mean Difference (Final Values) = -1.04, 60% CI 2-sided [-4.51 to 2.44], Standard Error of Mean 4.13
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0819, Mixed Models Analysis; Mean Difference (Final Values) = 5.63, 60% CI 2-sided [2.91 to 8.35], Standard Error of Mean 3.23
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.6103, Mixed Models Analysis; Mean Difference (Final Values) = -2.17, 60% CI 2-sided [-5.75 to 1.41], Standard Error of Mean 4.26
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.1168, Mixed Models Analysis; Mean Difference (Final Values) = 5.48, 60% CI 2-sided [2.54 to 8.41], Standard Error of Mean 3.49
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.3357, Mixed Models Analysis; Mean Difference (Final Values) = 4.26, 60% CI 2-sided [0.54 to 7.99], Standard Error of Mean 4.43
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0448, Mixed Models Analysis; Mean Difference (Final Values) = 7.42, 60% CI 2-sided [4.31 to 10.54], Standard Error of Mean 3.70
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.7642, Mixed Models Analysis; Mean Difference (Final Values) = 1.39, 60% CI 2-sided [-2.51 to 5.29], Standard Error of Mean 4.64
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.1295, Mixed Models Analysis; Mean Difference (Final Values) = 5.99, 60% CI 2-sided [2.67 to 9.32], Standard Error of Mean 3.95
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.6540, Mixed Models Analysis; Mean Difference (Final Values) = 2.13, 60% CI 2-sided [-1.87 to 6.13], Standard Error of Mean 4.75

15. Secondary Outcome: Least Squares Means of Total Serum Triglycerides (mg/dL) by Visit
Description: as for outcome 12
Time Frame: Month 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Population. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 49
mg/dL
  Month 15 | 177.33 (13.66) | 171.21 (13.94) | 167.38 (15.07)
  Month 18 | 181.92 (13.74) | 163.26 (13.97) | 145.05 (15.18)
  Month 24 (n=58,54,40) | 183.79 (13.93) | 162.80 (14.33) | 142.07 (16.23)
  Month 30 (n=52,37,26) | 182.49 (14.44) | 137.05 (16.28) | 178.56 (19.18)
  Month 36 (n=51,32,15) | 174.01 (14.73) | 145.27 (17.85) | 152.98 (24.50)
  Month 42 (n=44,31,15) | 178.93 (15.55) | 183.09 (18.64) | 148.62 (26.42)
  Month 48 (n=42,30,14) | 166.38 (16.08) | 196.86 (19.04) | 156.12 (27.76)
  Month 54 (n=41,31,13) | 163.57 (16.41) | 169.18 (19.07) | 178.24 (28.75)
  Month 60 (n=37,23,12) | 156.27 (17.10) | 173.20 (21.06) | 142.27 (29.89)
  Month 66 (n=34,20,11) | 165.83 (17.82) | 174.19 (22.54) | 158.73 (31.35)
  Month 72 (n=31,17,11) | 143.03 (18.63) | 165.10 (24.40) | 161.28 (31.94)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.7543, Mixed Models Analysis; Mean Difference (Final Values) = -6.11, 60% CI 2-sided [-22.55 to 10.33], Standard Error of Mean 19.53
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.6249, Mixed Models Analysis; Mean Difference (Final Values) = -9.95, 60% CI 2-sided [-27.07 to 7.17], Standard Error of Mean 20.33
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.3415, Mixed Models Analysis; Mean Difference (Final Values) = -18.66, 60% CI 2-sided [-35.17 to -2.15], Standard Error of Mean 19.61
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.0720, Mixed Models Analysis; Mean Difference (Final Values) = -36.86, 60% CI 2-sided [-54.10 to -19.63], Standard Error of Mean 20.47
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.2937, Mixed Models Analysis; Mean Difference (Final Values) = -21.00, 60% CI 2-sided [-37.83 to -4.17], Standard Error of Mean 19.99
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.0512, Mixed Models Analysis; Mean Difference (Final Values) = -41.72, 60% CI 2-sided [-59.72 to -23.73], Standard Error of Mean 21.38
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.0370, Mixed Models Analysis; Mean Difference (Final Values) = -45.43, 60% CI 2-sided [-63.75 to -27.11], Standard Error of Mean 21.76
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.8701, Mixed Models Analysis; Mean Difference (Final Values) = -3.92, 60% CI 2-sided [-24.13 to 16.28], Standard Error of Mean 24.00
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.2146, Mixed Models Analysis; Mean Difference (Final Values) = -28.75, 60% CI 2-sided [-48.24 to -9.25], Standard Error of Mean 23.15
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.4620, Mixed Models Analysis; Mean Difference (Final Values) = -21.03, 60% CI 2-sided [-45.09 to 3.03], Standard Error of Mean 28.58
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.8639, Mixed Models Analysis; Mean Difference (Final Values) = 4.16, 60% CI 2-sided [-16.28 to 24.60], Standard Error of Mean 24.28
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.3230, Mixed Models Analysis; Mean Difference (Final Values) = -30.30, 60% CI 2-sided [-56.11 to -4.50], Standard Error of Mean 30.65
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.2214, Mixed Models Analysis; Mean Difference (Final Values) = 30.49, 60% CI 2-sided [9.51 to 51.47], Standard Error of Mean 24.92
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.7492, Mixed Models Analysis; Mean Difference (Final Values) = -10.25, 60% CI 2-sided [-37.26 to 16.75], Standard Error of Mean 32.08
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.8236, Mixed Models Analysis; Mean Difference (Final Values) = 5.61, 60% CI 2-sided [-15.57 to 26.79], Standard Error of Mean 25.15
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.6578, Mixed Models Analysis; Mean Difference (Final Values) = 14.67, 60% CI 2-sided [-13.20 to 42.54], Standard Error of Mean 33.10
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.5326, Mixed Models Analysis; Mean Difference (Final Values) = 16.93, 60% CI 2-sided [-5.90 to 39.76], Standard Error of Mean 27.12
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.6845, Mixed Models Analysis; Mean Difference (Final Values) = -14.00, 60% CI 2-sided [-42.99 to 15.00], Standard Error of Mean 34.44
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.7713, Mixed Models Analysis; Mean Difference (Final Values) = 8.35, 60% CI 2-sided [-15.83 to 32.54], Standard Error of Mean 28.73
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.8438, Mixed Models Analysis; Mean Difference (Final Values) = -7.11, 60% CI 2-sided [-37.47 to 23.26], Standard Error of Mean 36.06
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.4724, Mixed Models Analysis; Mean Difference (Final Values) = 22.06, 60% CI 2-sided [-3.78 to 47.91], Standard Error of Mean 30.70
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.6218, Mixed Models Analysis; Mean Difference (Final Values) = 18.25, 60% CI 2-sided [-12.89 to 49.38], Standard Error of Mean 36.98

16. Secondary Outcome: Mean Absolute Neutrophil Counts (ANC) (Kelvin Per Millimeter Cubed [K/mm^3]) by Visit
Description: Follow-up visit included Month 74 visit for completers and 2-month postdose visit for early withdrawals.
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72 and Follow-up
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Mean (Standard Deviation); unit: k/mm^3
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 58 | 49
k/mm^3
  Month 15 (n=55,56,47) | 4.53 (1.82) | 4.23 (1.79) | 4.33 (1.76)
  Month 18 | 4.59 (1.98) | 3.87 (1.57) | 4.83 (2.84)
  Month 24 (n=54,52,39) | 4.62 (1.93) | 3.99 (1.43) | 4.38 (1.55)
  Month 30 (n=48,35,26) | 4.69 (1.91) | 3.48 (1.25) | 4.55 (1.71)
  Month 36 (n=51,30,15) | 4.48 (1.93) | 3.72 (1.41) | 4.62 (1.22)
  Month 42 (n=40,31,15) | 4.30 (1.80) | 3.90 (1.76) | 4.49 (0.81)
  Month 48 (n=41,30,13) | 3.86 (1.93) | 3.47 (1.58) | 3.86 (1.59)
  Month 54 (n=38,26,11) | 4.11 (1.78) | 3.42 (1.09) | 4.27 (1.52)
  Month 60 (n=37,20,11) | 4.30 (1.80) | 3.97 (1.57) | 4.01 (1.24)
  Month 66 (n=34,19,11) | 4.53 (1.85) | 3.86 (1.51) | 4.28 (1.21)
  Month 72 (n=31,17,11) | 4.33 (1.85) | 3.44 (1.12) | 4.73 (1.47)
  Follow-up (n=51,46,41) | 4.65 (1.77) | 3.75 (1.26) | 4.37 (1.97)

17. Secondary Outcome: Mean Hemoglobin (Hgb) (Grams Per Deciliter [g/dL]) by Visit
Description: Follow-up visit included Month 74 visit for completers and 2-month postdose visit for early withdrawals.
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72 and Follow-up
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 49
g/dL
  Month 15 (n=58,59,48) | 13.20 (1.78) | 13.14 (1.41) | 13.35 (1.65)
  Month 18 | 13.15 (1.71) | 13.31 (1.13) | 13.50 (1.86)
  Month 24 (n=57,54,41) | 13.35 (1.58) | 13.58 (1.25) | 13.58 (1.54)
  Month 30 (n=48,37,28) | 13.21 (1.66) | 13.66 (1.23) | 13.82 (1.60)
  Month 36 (n=52,32,15) | 13.30 (1.59) | 13.91 (1.08) | 13.44 (1.94)
  Month 42 (n=41,31,15) | 13.24 (1.60) | 13.99 (0.99) | 13.67 (1.70)
  Month 48 (n=42,31,13) | 13.05 (1.71) | 14.01 (1.18) | 13.28 (1.45)
  Month 54 (n=40,29,11) | 13.22 (1.53) | 13.98 (1.31) | 13.60 (1.54)
  Month 60 (n=37,20,12) | 13.29 (1.56) | 14.40 (1.24) | 13.41 (1.94)
  Month 66 (n=34,19,11) | 13.02 (1.88) | 14.62 (1.18) | 13.42 (2.14)
  Month 72 (n=31,17,11) | 13.10 (1.84) | 14.22 (1.56) | 13.23 (2.03)
  Follow-up (n=51,47,41) | 12.49 (2.04) | 13.23 (1.75) | 13.72 (2.09)

18. Secondary Outcome: Mean Glycosylated Hemoglobin (HBA1c) (Percent [%]) by Visit
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The normal range for the HbA1c test is between 4% and 5.6%. HbA1c levels between 5.7% and 6.4% indicate increased risk of diabetes and levels of 6.5% or higher indicate diabetes.
Time Frame: Months 24, 36, 48, 60, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 55 | 51 | 35
Percentage
  Month 24 | 6.35 (1.84) | 6.16 (1.53) | 6.37 (1.40)
  Month 36 (n=50,32,15) | 6.16 (1.39) | 5.92 (1.20) | 6.69 (2.31)
  Month 48 (n=43,31,14) | 6.15 (1.64) | 6.16 (1.88) | 6.59 (1.71)
  Month 60 (n=37,23,12) | 6.36 (1.94) | 6.26 (2.03) | 6.28 (1.88)
  Month 72 (n=31,16,11) | 6.52 (1.98) | 6.34 (1.57) | 6.33 (2.21)

19. Secondary Outcome: Least Squares Means of Fasting Serum Glucose Levels (mg/dL) by Visit
Description: Model contained treatment, visit and treatment by visit interaction as fixed effects and Baseline (predose in Study A3921030) as a covariate. A compund symmetry variance-covariance structure was used.
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Population. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 49
mg/dL
  Month 15 (n=59,58,49) | 104.42 (5.56) | 102.10 (5.66) | 107.18 (6.13)
  Month 18 | 113.01 (5.57) | 106.17 (5.63) | 107.56 (6.13)
  Month 24 (n=58,54,41) | 112.23 (5.60) | 107.81 (5.79) | 102.47 (6.50)
  Month 30 (n=50,38,27) | 105.27 (5.87) | 108.01 (6.53) | 107.70 (7.55)
  Month 36 (n=51,32,15) | 95.88 (5.84) | 106.27 (6.95) | 106.03 (9.55)
  Month 42 (n=44,31,15) | 107.10 (6.14) | 114.43 (7.03) | 94.16 (9.55)
  Month 48 (n=42,30,14) | 101.14 (6.23) | 109.86 (7.12) | 104.07 (9.83)
  Month 54 (n=41,31,13) | 114.50 (6.29) | 110.62 (7.04) | 127.38 (10.13)
  Month 60 (n=37,23,12) | 109.75 (6.52) | 106.64 (7.88) | 107.49 (10.49)
  Month 66 (n=34,20,11) | 104.42 (6.72) | 103.25 (8.33) | 108.55 (10.88)
  Month 72 (n=30,17,11) | 107.01 (7.04) | 105.22 (8.89) | 99.82 (10.88)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.7693, Mixed Models Analysis; Mean Difference (Final Values) = -2.33, 60% CI 2-sided [-9.01 to 4.35], Standard Error of Mean 7.93
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.7396, Mixed Models Analysis; Mean Difference (Final Values) = 2.75, 60% CI 2-sided [-4.22 to 9.73], Standard Error of Mean 8.28
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.3881, Mixed Models Analysis; Mean Difference (Final Values) = -6.84, 60% CI 2-sided [-13.51 to -0.17], Standard Error of Mean 7.92
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.5114, Mixed Models Analysis; Mean Difference (Final Values) = -5.44, 60% CI 2-sided [-12.42 to 1.53], Standard Error of Mean 8.28
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.5829, Mixed Models Analysis; Mean Difference (Final Values) = -4.43, 60% CI 2-sided [-11.21 to 2.36], Standard Error of Mean 8.06
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.2559, Mixed Models Analysis; Mean Difference (Final Values) = -9.76, 60% CI 2-sided [-16.99 to -2.53], Standard Error of Mean 8.58
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.7548, Mixed Models Analysis; Mean Difference (Final Values) = 2.74, 60% CI 2-sided [-4.65 to 10.14], Standard Error of Mean 8.78
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Match 30; Test type: Superiority or Other; p = 0.7998, Mixed Models Analysis; Mean Difference (Final Values) = 2.43, 60% CI 2-sided [-5.63 to 10.49], Standard Error of Mean 9.57
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.2531, Mixed Models Analysis; Mean Difference (Final Values) = 10.39, 60% CI 2-sided [2.74 to 18.03], Standard Error of Mean 9.08
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.3650, Mixed Models Analysis; Mean Difference (Final Values) = 10.14, 60% CI 2-sided [0.72 to 19.57], Standard Error of Mean 11.20
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.4328, Mixed Models Analysis; Mean Difference (Final Values) = 7.33, 60% CI 2-sided [-0.53 to 15.19], Standard Error of Mean 9.34
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.2547, Mixed Models Analysis; Mean Difference (Final Values) = -12.94, 60% CI 2-sided [-22.50 to -3.38], Standard Error of Mean 11.35
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.3572, Mixed Models Analysis; Mean Difference (Final Values) = 8.72, 60% CI 2-sided [0.75 to 16.69], Standard Error of Mean 9.46
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.8009, Mixed Models Analysis; Mean Difference (Final Values) = 2.94, 60% CI 2-sided [-6.86 to 12.74], Standard Error of Mean 11.64
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.6814, Mixed Models Analysis; Mean Difference (Final Values) = -3.88, 60% CI 2-sided [-11.82 to 4.07], Standard Error of Mean 9.44
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.2803, Mixed Models Analysis; Mean Difference (Final Values) = 12.88, 60% CI 2-sided [2.84 to 22.93], Standard Error of Mean 11.93
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.7613, Mixed Models Analysis; Mean Difference (Final Values) = -3.11, 60% CI 2-sided [-11.72 to 5.50], Standard Error of Mean 10.23
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.8554, Mixed Models Analysis; Mean Difference (Final Values) = -2.25, 60% CI 2-sided [-12.65 to 8.15], Standard Error of Mean 12.35
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.9132, Mixed Models Analysis; Mean Difference (Final Values) = -1.17, 60% CI 2-sided [-10.18 to 7.84], Standard Error of Mean 10.70
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.7465, Mixed Models Analysis; Mean Difference (Final Values) = 4.14, 60% CI 2-sided [-6.63 to 14.90], Standard Error of Mean 12.79
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.8747, Mixed Models Analysis; Mean Difference (Final Values) = -1.79, 60% CI 2-sided [-11.34 to 7.76], Standard Error of Mean 11.34
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.5793, Mixed Models Analysis; Mean Difference (Final Values) = -7.19, 60% CI 2-sided [-18.10 to 3.72], Standard Error of Mean 12.96

20. Secondary Outcome: Percentage of Participants by Proteinuria Category by Visit
Description: Proteinuria was defined as the presence of an excess of serum proteins in the urine. Normal value of proteinuria is below 0.15 grams per 24 hours (g/24 hr). Follow-up visit included Month 74 visit for completers and 2-month postdose visit for early withdrawals.
Time Frame: Months 24, 36, 48, 60, 72 and Follow-up
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 51 | 47 | 36
Percentage of Participants
  Month 24: >200 mg/day | 15.7 | 27.7 | 19.4
  Month 24: >500 mg/day | 3.9 | 6.4 | 8.3
  Month 24: >1500 mg/day | 2.0 | 2.1 | 5.6
  Month 24: >500 Increase from Baseline | 2.0 | 0 | 0
  Month 36: >200 mg/day (n=42,30,13) | 14.3 | 26.7 | 15.4
  Month 36: >500 mg/day (n=42,30,13) | 2.4 | 3.3 | 0
  Month 36: >1500 mg/day (n=42,30,13) | 2.4 | 3.3 | 0
  Month 36: >500 Increase from Baseline (n=42,30,13) | 0 | 0 | 0
  Month 48: >200 mg/day (n=36,29,12) | 16.7 | 31.0 | 0
  Month 48: >500 mg/day (n=36,29,12) | 5.6 | 17.2 | 0
  Month 48: >1500 mg/day (n=36,29,12) | 2.8 | 6.9 | 0
  Month 48: >500 Increase in Baseline (n=36,29,12) | 0 | 3.4 | 0
  Month 60: >200 mg/day (n=29,20,10) | 10.3 | 20.0 | 10.0
  Month 60: >500 mg/day (n=29,20,10) | 10.3 | 15.0 | 0
  Month 60: >1500 mg/day (n=29,20,10) | 3.4 | 5.0 | 0
  Month 60: >500 Increase in Baseline (n=29,20,10) | 0 | 5.0 | 0
  Month 72: >200 mg/day (n=22,15,9) | 9.1 | 20.0 | 22.2
  Month 72: >500 mg/day (n=22,15,9) | 4.5 | 20.0 | 11.1
  Month 72: >1500 mg/day (n=22,15,9) | 0 | 13.3 | 0
  Month 72: >500 Increase in Baseline (n=22,15,9) | 0 | 0 | 11.1
  Follow-up: >200 mg/day (n=46,34,39) | 13.0 | 17.6 | 20.5
  Follow-up: >500 mg/day (n=46,34,39) | 6.5 | 8.8 | 5.1
  Follow-up: >1500 mg/day (n=46,34,39) | 2.2 | 5.9 | 2.6
  Follow-up: >500 Increase in Baseline (n=46,34,39) | 0 | 0 | 2.6

21. Secondary Outcome: Least Square Means of Estimated GFR Calculated Using the Nankivell Equation by Visit
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated using Nankivell formula, where:
  Creatinine clearance (mL/min) = 6.7/serum creatinine (millimols per litre [mmol/L]) - serum urea (mmol/dL)/2 + actual body weight (kilograms [kg])/4 - 100/Height (metres [m])^2 + (35 for male or 25 for female).
  A normal GFR for adults is > 90 mL/min. Lower values indicate poor kidney function. A GFR <15 is consistent with kidney failure.
  Model contained treatment, visit and treatment by visit interaction as fixed effects. An unstructured variance-covariance structure was used.
Time Frame: Month 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: minutes per milliliter (min/mL)
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 50
minutes per milliliter (min/mL)
  Month 15 | 69.57 (1.95) | 82.33 (2.00) | 82.96 (2.13)
  Month 18 | 70.93 (2.09) | 82.41 (2.15) | 82.91 (2.28)
  Month 24 (n=58,54,41) | 69.78 (2.09) | 82.63 (2.15) | 83.49 (2.32)
  Month 30 (n=51,37,27) | 68.41 (2.28) | 84.27 (2.46) | 82.02 (2.73)
  Month 36 (n=51,32,15) | 68.94 (2.44) | 81.10 (2.66) | 81.50 (3.14)
  Month 42 (n=44,31,15) | 68.82 (2.29) | 81.24 (2.49) | 77.81 (2.98)
  Month 48 (n=42,30,14) | 67.68 (2.54) | 80.08 (2.79) | 75.28 (3.46)
  Month 54 (n=41,31,13) | 65.59 (2.69) | 79.63 (2.98) | 75.82 (3.88)
  Month 60 (n=37,24,12) | 70.08 (2.46) | 77.80 (2.77) | 74.19 (3.51)
  Month 66 (n=34,20,11) | 68.99 (2.80) | 76.74 (3.17) | 75.01 (4.01)
  Month 72 (n=30,17,11) | 68.65 (3.39) | 81.68 (4.01) | 72.92 (5.10)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 12.76, 60% CI 2-sided [10.40 to 15.11], Standard Error of Mean 2.79
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 13.39, 60% CI 2-sided [10.96 to 15.82], Standard Error of Mean 2.88
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 11.48, 60% CI 2-sided [8.95 to 14.00], Standard Error of Mean 3.00
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 11.98, 60% CI 2-sided [9.37 to 14.59], Standard Error of Mean 3.09
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 12.86, 60% CI 2-sided [10.32 to 15.39], Standard Error of Mean 3.00
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 13.71, 60% CI 2-sided [11.08 to 16.35], Standard Error of Mean 3.12
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 15.86, 60% CI 2-sided [13.03 to 18.69], Standard Error of Mean 3.35
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 13.61, 60% CI 2-sided [10.61 to 16.61], Standard Error of Mean 3.56
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = 12.17, 60% CI 2-sided [9.12 to 15.21], Standard Error of Mean 3.61
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; Mean Difference (Final Values) = 12.56, 60% CI 2-sided [9.20 to 15.92], Standard Error of Mean 3.98
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 12.42, 60% CI 2-sided [9.56 to 15.27], Standard Error of Mean 3.38
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.0182, Mixed Models Analysis; Mean Difference (Final Values) = 8.99, 60% CI 2-sided [5.81 to 12.16], Standard Error of Mean 3.76
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Mean Difference (Final Values) = 12.40, 60% CI 2-sided [9.22 to 15.58], Standard Error of Mean 3.77
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.0782, Mixed Models Analysis; Mean Difference (Final Values) = 7.60, 60% CI 2-sided [3.99 to 11.22], Standard Error of Mean 4.29
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = 14.04, 60% CI 2-sided [10.64 to 17.43], Standard Error of Mean 4.02
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.0322, Mixed Models Analysis; Mean Difference (Final Values) = 10.23, 60% CI 2-sided [6.24 to 14.22], Standard Error of Mean 4.72
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0399, Mixed Models Analysis; Mean Difference (Final Values) = 7.72, 60% CI 2-sided [4.59 to 10.86], Standard Error of Mean 3.70
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.3391, Mixed Models Analysis; Mean Difference (Final Values) = 4.11, 60% CI 2-sided [0.49 to 7.73], Standard Error of Mean 4.28
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0702, Mixed Models Analysis; Mean Difference (Final Values) = 7.75, 60% CI 2-sided [4.17 to 11.33], Standard Error of Mean 4.23
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.2210, Mixed Models Analysis; Mean Difference (Final Values) = 6.02, 60% CI 2-sided [1.89 to 10.15], Standard Error of Mean 4.89
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0150, Mixed Models Analysis; Mean Difference (Final Values) = 13.03, 60% CI 2-sided [8.59 to 17.46], Standard Error of Mean 5.25
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.4875, Mixed Models Analysis; Mean Difference (Final Values) = 4.27, 60% CI 2-sided [-0.91 to 9.45], Standard Error of Mean 6.13

22. Secondary Outcome: Least Squares Means of Estimated GFR Calculated Using the Cockcroft-Gault Equation by Visit
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR (mL/min) was calculated using Cockcroft-Gault equation. GFR by Cockcroft-Gault equation= body weight (kg)*(140 minus age in years) divided by (72*serum creatinine [mg/dL]). For females value obtained was multiplied by 0.85. A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
  Model contained treatment, visit and treatment by visit interaction as fixed effects. An unstructured variance-covariance structure was used.
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: min/mL
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 59 | 59 | 50
min/mL
  Month 15 | 72.74 (3.02) | 87.22 (3.10) | 87.67 (3.29)
  Month 18 | 73.56 (3.14) | 87.52 (3.23) | 87.12 (3.42)
  Month 24 (n=58,54,42) | 72.70 (3.28) | 87.72 (3.39) | 87.62 (3.62)
  Month 30 (n=51,38,29) | 70.70 (3.48) | 89.24 (3.68) | 87.15 (3.99)
  Month 36 (n=51,32,15) | 70.71 (3.75) | 85.91 (4.04) | 85.64 (4.68)
  Month 42 (n=44,31,15) | 69.63 (3.48) | 85.95 (3.76) | 81.88 (4.45)
  Month 48 (n=42,30,14) | 67.63 (3.81) | 83.96 (4.15) | 77.42 (5.03)
  Month 54 (n=41,31,13) | 65.81 (3.85) | 82.78 (4.20) | 77.60 (5.26)
  Month 60 (n=37,24,12) | 70.52 (3.92) | 78.54 (4.43) | 74.18 (5.63)
  Month 66 (n=34,20,11) | 69.09 (3.81) | 79.09 (4.21) | 74.52 (5.11)
  Month 72 (n=30,17,11) | 68.34 (4.44) | 85.50 (5.11) | 73.05 (6.45)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = 14.48, 60% CI 2-sided [10.83 to 18.13], Standard Error of Mean 4.33
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = 14.93, 60% CI 2-sided [11.16 to 18.70], Standard Error of Mean 4.47
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; Mean Difference (Final Values) = 13.96, 60% CI 2-sided [10.16 to 17.76], Standard Error of Mean 4.50
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; Mean Difference (Final Values) = 13.57, 60% CI 2-sided [9.65 to 17.48], Standard Error of Mean 4.64
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; Mean Difference (Final Values) = 15.02, 60% CI 2-sided [11.04 to 19.00], Standard Error of Mean 4.72
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; Mean Difference (Final Values) = 14.93, 60% CI 2-sided [10.81 to 19.04], Standard Error of Mean 4.88
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 18.54, 60% CI 2-sided [14.27 to 22.81], Standard Error of Mean 5.06
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = 16.45, 60% CI 2-sided [11.99 to 20.91], Standard Error of Mean 5.29
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; Mean Difference (Final Values) = 15.19, 60% CI 2-sided [10.55 to 19.84], Standard Error of Mean 5.51
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.0137, Mixed Models Analysis; Mean Difference (Final Values) = 14.93, 60% CI 2-sided [9.87 to 19.99], Standard Error of Mean 6.00
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = 16.32, 60% CI 2-sided [11.99 to 20.64], Standard Error of Mean 5.12
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.0316, Mixed Models Analysis; Mean Difference (Final Values) = 12.24, 60% CI 2-sided [7.47 to 17.01], Standard Error of Mean 5.65
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0043, Mixed Models Analysis; Mean Difference (Final Values) = 16.33, 60% CI 2-sided [11.57 to 21.09], Standard Error of Mean 5.64
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.1226, Mixed Models Analysis; Mean Difference (Final Values) = 9.80, 60% CI 2-sided [4.47 to 15.12], Standard Error of Mean 6.31
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; Mean Difference (Final Values) = 16.97, 60% CI 2-sided [12.17 to 21.78], Standard Error of Mean 5.70
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.0724, Mixed Models Analysis; Mean Difference (Final Values) = 11.79, 60% CI 2-sided [6.29 to 17.29], Standard Error of Mean 6.52
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.1782, Mixed Models Analysis; Mean Difference (Final Values) = 8.03, 60% CI 2-sided [3.02 to 13.03], Standard Error of Mean 5.92
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.5947, Mixed Models Analysis; Mean Difference (Final Values) = 3.66, 60% CI 2-sided [-2.14 to 9.46], Standard Error of Mean 6.86
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0810, Mixed Models Analysis; Mean Difference (Final Values) = 9.99, 60% CI 2-sided [5.20 to 14.79], Standard Error of Mean 5.68
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.3965, Mixed Models Analysis; Mean Difference (Final Values) = 5.42, 60% CI 2-sided [0.04 to 10.81], Standard Error of Mean 6.38
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0128, Mixed Models Analysis; Mean Difference (Final Values) = 17.16, 60% CI 2-sided [11.44 to 22.88], Standard Error of Mean 6.77
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.5487, Mixed Models Analysis; Mean Difference (Final Values) = 4.71, 60% CI 2-sided [-1.91 to 11.33], Standard Error of Mean 7.83

23. Secondary Outcome: Least Squares Means of Estimated GFR (eGFR) (mL/Min/1.73 Square Meter [m^2]) Calculated by the Modification of Diet in Renal Disease (MDRD) Equation With Last Observation Carried Forward (LOCF) Plus Imputation (eGFR=0 for Graft Loss/Death) by Visit
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using MDRD equation. GFR (mL/min/1.73 m^2) by MDRD equation = 170 * (serum creatinine [mg/dL])^(-0.999) * (age in years)^(-0.176) * (0.762 if female) * (1.18 if black) * (blood urea nitrogen concentration [mg/dL])^(-0.170) * (serum albumin concentration [g/dL])^(0.318). A normal GFR is >90 mL/min/1.73 m^2, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min/1.73 m^2 indicated kidney failure.
  Model contained treatment, visit and treatment by visit interaction as fixed effects. An unstructured variance-covariance structure was used.
Time Frame: Months 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72
Population: Safety Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 64 | 60 | 54
mL/min/1.73m^2
  Month 15 | 56.25 (1.99) | 72.12 (2.06) | 70.22 (2.17)
  Month 18 | 58.13 (2.32) | 71.66 (2.39) | 69.69 (2.52)
  Month 24 | 56.30 (2.40) | 71.93 (2.47) | 68.20 (2.61)
  Month 30 | 53.82 (2.69) | 73.10 (2.78) | 64.44 (2.93)
  Month 36 | 54.37 (3.00) | 69.09 (3.10) | 63.27 (3.26)
  Month 42 | 53.59 (2.96) | 68.29 (3.05) | 62.14 (3.22)
  Month 48 | 51.69 (3.23) | 65.27 (3.34) | 60.81 (3.52)
  Month 54 | 48.64 (3.29) | 65.25 (3.40) | 60.79 (3.59)
  Month 60 | 50.43 (3.30) | 63.82 (3.41) | 59.20 (3.59)
  Month 66 | 49.70 (3.34) | 63.33 (3.45) | 59.47 (3.63)
  Month 72 | 49.62 (3.51) | 64.27 (3.62) | 59.21 (3.82)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 15; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 15.87, 60% CI 2-sided [13.46 to 18.29], Standard Error of Mean 2.86
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 15; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 13.97, 60% CI 2-sided [11.49 to 16.46], Standard Error of Mean 2.95
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 18; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 13.53, 60% CI 2-sided [10.71 to 16.34], Standard Error of Mean 3.33
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 18; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = 11.56, 60% CI 2-sided [8.67 to 14.45], Standard Error of Mean 3.43
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 15.63, 60% CI 2-sided [12.72 to 18.53], Standard Error of Mean 3.44
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = 11.89, 60% CI 2-sided [8.91 to 14.88], Standard Error of Mean 3.54
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 30; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 19.29, 60% CI 2-sided [16.03 to 22.55], Standard Error of Mean 3.86
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 30; Test type: Superiority or Other; p = 0.0082, Mixed Models Analysis; Mean Difference (Final Values) = 10.63, 60% CI 2-sided [7.27 to 13.98], Standard Error of Mean 3.97
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = 14.72, 60% CI 2-sided [11.09 to 18.36], Standard Error of Mean 4.31
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36; Test type: Superiority or Other; p = 0.0462, Mixed Models Analysis; Mean Difference (Final Values) = 8.90, 60% CI 2-sided [5.16 to 12.64], Standard Error of Mean 4.43
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 42; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = 14.70, 60% CI 2-sided [11.11 to 18.28], Standard Error of Mean 4.25
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 42; Test type: Superiority or Other; p = 0.0519, Mixed Models Analysis; Mean Difference (Final Values) = 8.55, 60% CI 2-sided [4.87 to 12.24], Standard Error of Mean 4.37
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 48; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; Mean Difference (Final Values) = 13.58, 60% CI 2-sided [9.66 to 17.50], Standard Error of Mean 4.65
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 48; Test type: Superiority or Other; p = 0.0580, Mixed Models Analysis; Mean Difference (Final Values) = 9.12, 60% CI 2-sided [5.09 to 13.15], Standard Error of Mean 4.78
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 54; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = 16.61, 60% CI 2-sided [12.62 to 20.61], Standard Error of Mean 4.74
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 54; Test type: Superiority or Other; p = 0.0136, Mixed Models Analysis; Mean Difference (Final Values) = 12.15, 60% CI 2-sided [8.04 to 16.26], Standard Error of Mean 4.87
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 60; Test type: Superiority or Other; p = 0.0053, Mixed Models Analysis; Mean Difference (Final Values) = 13.39, 60% CI 2-sided [9.39 to 17.39], Standard Error of Mean 4.74
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 60; Test type: Superiority or Other; p = 0.0736, Mixed Models Analysis; Mean Difference (Final Values) = 8.77, 60% CI 2-sided [4.66 to 12.88], Standard Error of Mean 4.87
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 66; Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis; Mean Difference (Final Values) = 13.63, 60% CI 2-sided [9.58 to 17.67], Standard Error of Mean 4.80
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 66; Test type: Superiority or Other; p = 0.0491, Mixed Models Analysis; Mean Difference (Final Values) = 9.77, 60% CI 2-sided [5.61 to 13.93], Standard Error of Mean 4.93
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 72; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; Mean Difference (Final Values) = 14.66, 60% CI 2-sided [10.40 to 18.91], Standard Error of Mean 5.04
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 72; Test type: Superiority or Other; p = 0.0660, Mixed Models Analysis; Mean Difference (Final Values) = 9.59, 60% CI 2-sided [5.22 to 13.97], Standard Error of Mean 5.19

24. Secondary Outcome: Least Squares Means of Short Form 36 Version 2 (SF-36 V2) Component and Domain Scores at Months 24 and 36
Description: SF-36 v2 is a self-administered 36-item generic health status measure with 8 general health concepts which are the weighted sums of the questions in their section: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health. Each scale is transformed into a 0 (minimum) to 100 (maximum) scale on the assumption each question carries equal weight. These concepts were also summarized into 2 summary scores; Physical Component Summary and Mental Component Summary (both a 0-100 scale). The 8 subscales, 2 summary scores and transition Question 2 (TR Scale, measured on a scale of 1 [minimum] to 5 [maximum]) were subjected to analysis. Higher domain, summary scores, and TR scale scores indicate better health status. Model contained treatment, visit and treatment by visit interaction as fixed effects and Baseline (predose in Study A3921030) as a covariate. First-order autoregressive variance-covariance structure was used.
Time Frame: Months 24, 36
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 41 | 33 | 24
Score on a scale
  Month 24: Physical Functioning | 49.04 (1.16) | 47.00 (1.29) | 45.47 (1.49)
  Month 24: Role Physical | 46.36 (1.41) | 47.72 (1.56) | 44.40 (1.82)
  Month 24: Bodily Pain | 51.37 (1.42) | 51.66 (1.58) | 51.47 (1.84)
  Month 24: General Health | 46.51 (1.19) | 48.25 (1.32) | 47.60 (1.54)
  Month 24: Vitality | 53.31 (1.25) | 53.27 (1.39) | 55.07 (1.64)
  Month 24: Social Functioning | 49.55 (1.33) | 49.41 (1.47) | 49.95 (1.74)
  Month 24: Role Emotional | 44.65 (1.55) | 48.47 (1.72) | 44.17 (2.01)
  Month 24: Mental Health | 49.52 (1.35) | 47.83 (1.50) | 53.08 (1.76)
  Month 24: TR Scale Score | 2.63 (0.10) | 2.85 (0.12) | 2.86 (0.14)
  Month 24: Physical Component Summary | 49.00 (1.13) | 48.99 (1.25) | 46.57 (1.45)
  Month 24: Mental Component Summary | 48.65 (1.29) | 49.62 (1.43) | 51.92 (1.68)
  Month 36 (n=35,21,10): Physical Functioning | 48.62 (1.25) | 46.97 (1.60) | 46.18 (2.27)
  Month 36 (n=35,21,10): Role Physical | 48.00 (1.52) | 48.52 (1.94) | 46.00 (2.79)
  Month 36 (n=35,21,10): Bodily Pain | 50.57 (1.54) | 52.66 (1.97) | 50.19 (2.84)
  Month 36 (n=35,21,10): General Health | 46.06 (1.29) | 47.83 (1.63) | 47.02 (2.32)
  Month 36 (n=35,21,10): Vitality | 53.01 (1.35) | 54.45 (1.73) | 57.43 (2.50)
  Month 36 (n=35,21,10): Social Functioning | 48.96 (1.44) | 51.43 (1.84) | 48.33 (2.65)
  Month 36 (n=35,21,10): Role Emotional | 46.35 (1.68) | 51.97 (2.15) | 47.58 (3.09)
  Month 36 (n=35,21,10): Mental health | 50.21 (1.46) | 51.84 (1.86) | 50.59 (2.68)
  Month 36 (n=35,21,10): TR Scale Score | 2.46 (0.11) | 2.65 (0.14) | 2.83 (0.21)
  Month 36 (n=35,21,10): Physical Component Summary | 48.55 (1.22) | 48.00 (1.55) | 47.07 (2.21)
  Month 36 (n=35,21,10): Mental Component Summary | 49.45 (1.39) | 53.50 (1.77) | 52.32 (2.55)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Physical Functioning; Test type: Superiority or Other; p = 0.2393, Mixed Models Analysis; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-5.45 to 1.36], Standard Error of Mean 1.73
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Physical Functioning; Test type: Superiority or Other; p = 0.0595, Mixed Models Analysis; Mean Difference (Final Values) = -3.57, 95% CI 2-sided [-7.29 to 0.14], Standard Error of Mean 1.89
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Role Physical; Test type: Superiority or Other; p = 0.5182, Mixed Models Analysis; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [-2.77 to 5.49], Standard Error of Mean 2.10
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Role Physical; Test type: Superiority or Other; p = 0.3938, Mixed Models Analysis; Mean Difference (Final Values) = -1.96, 95% CI 2-sided [-6.49 to 2.56], Standard Error of Mean 2.30
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Bodily Pain; Test type: Superiority or Other; p = 0.8932, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-3.89 to 4.46], Standard Error of Mean 2.12
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Bodily Pain; Test type: Superiority or Other; p = 0.9673, Mixed Models Analysis; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-4.48 to 4.67], Standard Error of Mean 2.33
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: General Health; Test type: Superiority or Other; p = 0.3290, Mixed Models Analysis; Mean Difference (Final Values) = 1.74, 95% CI 2-sided [-1.76 to 5.23], Standard Error of Mean 1.78
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: General Health; Test type: Superiority or Other; p = 0.5780, Mixed Models Analysis; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-2.75 to 4.92], Standard Error of Mean 1.95
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Vitality; Test type: Superiority or Other; p = 0.9799, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-3.72 to 3.62], Standard Error of Mean 1.87
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Vitality; Test type: Superiority or Other; p = 0.3960, Mixed Models Analysis; Mean Difference (Final Values) = 1.76, 95% CI 2-sided [-2.31 to 5.83], Standard Error of Mean 2.07
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Social Functioning; Test type: Superiority or Other; p = 0.9400, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-4.05 to 3.75], Standard Error of Mean 1.98
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Social Functioning; Test type: Superiority or Other; p = 0.8583, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-3.94 to 4.72], Standard Error of Mean 2.20
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Role Emotional; Test type: Superiority or Other; p = 0.0997, Mixed Models Analysis; Mean Difference (Final Values) = 3.82, 95% CI 2-sided [-0.73 to 8.37], Standard Error of Mean 2.31
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Role Emotional; Test type: Superiority or Other; p = 0.8520, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-5.47 to 4.52], Standard Error of Mean 2.54
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Mental Health; Test type: Superiority or Other; p = 0.4023, Mixed Models Analysis; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-5.64 to 2.27], Standard Error of Mean 2.01
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Mental Health; Test type: Superiority or Other; p = 0.1092, Mixed Models Analysis; Mean Difference (Final Values) = 3.56, 95% CI 2-sided [-0.80 to 7.92], Standard Error of Mean 2.22
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: TR Scale Score; Test type: Superiority or Other; p = 0.1754, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.10 to 0.52], Standard Error of Mean 0.16
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: TR Scale Score; Test type: Superiority or Other; p = 0.1802, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.11 to 0.57], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Physical Component Summary; Test type: Superiority or Other; p = 0.9966, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-3.31 to 3.29], Standard Error of Mean 1.68
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Physical Component Summary; Test type: Superiority or Other; p = 0.1880, Mixed Models Analysis; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-6.04 to 1.19], Standard Error of Mean 1.84
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24: Mental Component Summary; Test type: Superiority or Other; p = 0.6154, Mixed Models Analysis; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-2.81 to 4.73], Standard Error of Mean 1.92
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24: Mental Component Summary; Test type: Superiority or Other; p = 0.1248, Mixed Models Analysis; Mean Difference (Final Values) = 3.26, 95% CI 2-sided [-0.91 to 7.43], Standard Error of Mean 2.12
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Physical Functioning; Test type: Superiority or Other; p = 0.4174, Mixed Models Analysis; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-5.63 to 2.34], Standard Error of Mean 2.03
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Physical Functioning; Test type: Superiority or Other; p = 0.3486, Mixed Models Analysis; Mean Difference (Final Values) = -2.44, 95% CI 2-sided [-7.54 to 2.66], Standard Error of Mean 2.60
Statistical Analysis 25: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Role Physical; Test type: Superiority or Other; p = 0.8335, Mixed Models Analysis; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-4.33 to 5.37], Standard Error of Mean 2.47
Statistical Analysis 26: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Role Physical; Test type: Superiority or Other; p = 0.5291, Mixed Models Analysis; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-8.24 to 4.24], Standard Error of Mean 3.18
Statistical Analysis 27: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Bodily Pain; Test type: Superiority or Other; p = 0.4033, Mixed Models Analysis; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [-2.82 to 7.00], Standard Error of Mean 2.50
Statistical Analysis 28: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Bodily Pain; Test type: Superiority or Other; p = 0.9078, Mixed Models Analysis; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-6.74 to 5.99], Standard Error of Mean 3.24
Statistical Analysis 29: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: General Health; Test type: Superiority or Other; p = 0.3947, Mixed Models Analysis; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [-2.31 to 5.86], Standard Error of Mean 2.08
Statistical Analysis 30: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: General Health; Test type: Superiority or Other; p = 0.7165, Mixed Models Analysis; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-4.26 to 6.20], Standard Error of Mean 2.66
Statistical Analysis 31: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Vitality; Test type: Superiority or Other; p = 0.5112, Mixed Models Analysis; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-2.87 to 5.75], Standard Error of Mean 2.19
Statistical Analysis 32: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Vitality; Test type: Superiority or Other; p = 0.1218, Mixed Models Analysis; Mean Difference (Final Values) = 4.43, 95% CI 2-sided [-1.18 to 10.04], Standard Error of Mean 2.86
Statistical Analysis 33: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Social Functioning; Test type: Superiority or Other; p = 0.2895, Mixed Models Analysis; Mean Difference (Final Values) = 2.47, 95% CI 2-sided [-2.11 to 7.05], Standard Error of Mean 2.33
Statistical Analysis 34: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Social Functioning; Test type: Superiority or Other; p = 0.8349, Mixed Models Analysis; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-6.58 to 5.32], Standard Error of Mean 3.03
Statistical Analysis 35: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Role Emotional; Test type: Superiority or Other; p = 0.0393, Mixed Models Analysis; Mean Difference (Final Values) = 5.62, 95% CI 2-sided [0.28 to 10.97], Standard Error of Mean 2.72
Statistical Analysis 36: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Role Emotional; Test type: Superiority or Other; p = 0.7266, Mixed Models Analysis; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-5.69 to 8.16], Standard Error of Mean 3.52
Statistical Analysis 37: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Mental Health; Test type: Superiority or Other; p = 0.4916, Mixed Models Analysis; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [-3.02 to 6.27], Standard Error of Mean 2.36
Statistical Analysis 38: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Mental Health; Test type: Superiority or Other; p = 0.9008, Mixed Models Analysis; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-5.62 to 6.38], Standard Error of Mean 3.05
Statistical Analysis 39: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: TR Scale Score; Test type: Superiority or Other; p = 0.2965, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.17 to 0.55], Standard Error of Mean 0.18
Statistical Analysis 40: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: TR Scale Score; Test type: Superiority or Other; p = 0.1147, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.09 to 0.84], Standard Error of Mean 0.24
Statistical Analysis 41: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Physical Component Summary; Test type: Superiority or Other; p = 0.7786, Mixed Models Analysis; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-4.42 to 3.31], Standard Error of Mean 1.97
Statistical Analysis 42: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Physical Component Summary; Test type: Superiority or Other; p = 0.5582, Mixed Models Analysis; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-6.45 to 3.49], Standard Error of Mean 2.53
Statistical Analysis 43: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36: Mental Component Summary; Test type: Superiority or Other; p = 0.0727, Mixed Models Analysis; Mean Difference (Final Values) = 4.05, 95% CI 2-sided [-0.37 to 8.47], Standard Error of Mean 2.25
Statistical Analysis 44: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36: Mental Component Summary; Test type: Superiority or Other; p = 0.3264, Mixed Models Analysis; Mean Difference (Final Values) = 2.86, 95% CI 2-sided [-2.86 to 8.59], Standard Error of Mean 2.91

25. Secondary Outcome: Least Squares Means of End-Stage Renal Disease (ESRD) Symptom Checklist (SCL) -Transplantation Modules at Months 24 and 36
Description: ESRD-SCL: a 43-item disease specific self-administered questionnaire. Participants' rated the question "At the moment,how much do you suffer?" for each item on a 5 point scale, range (Ra) from 0 (not at all) to 4 (extremely). Consisted of 6 subscales: Cardiac and Renal (CR) dysfunction; Ra 0 to 28, Increased(In) Growth of Gum and Hair (IGGH); Ra 0 to 20, Limited Cognitive Capacity (LCC); Ra 0 to 32, Limited Physical Capacity (LPC); Ra 0 to 40, Side Effects (SEs) of Corticosteroids; Ra 0 to 20, Transplantation Associated Psychological Distress (TAPD); Ra 0 to 32. Total Score: 0 to 172, higher scores indicate greater dysfunction.
  Model contained treatment, visit and treatment by visit interaction as fixed effects and Baseline (predose in Study A3921030) as a covariate. A first-order autoregressive variance-covariance structure was used.
Time Frame: Months 24, 36
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 40 | 34 | 23
Score on a scale
  Month 24 Limited Physical Capacity (n=40,33,23) | 0.59 (0.07) | 0.70 (0.08) | 0.71 (0.10)
  Month 24 Limited Cognitive Capacity | 0.63 (0.08) | 0.71 (0.08) | 0.75 (0.10)
  Month 24 CR Dysfunction (n=40,33,23) | 0.63 (0.07) | 0.58 (0.08) | 0.53 (0.10)
  Month 24 SE of Corticosteroids (40, 33, 23) | 0.42 (0.08) | 0.57 (0.09) | 0.60 (0.11)
  Month 24 IGGH (n=40,33,23) | 0.54 (0.07) | 0.19 (0.08) | 0.17 (0.09)
  Month 24 TAPD | 0.61 (0.08) | 0.77 (0.09) | 0.63 (0.11)
  Month 24 Global Score (n=40,33,23) | 0.58 (0.06) | 0.62 (0.06) | 0.59 (0.07)
  Month 36 Limited Physical Capacity (n=33,21,8) | 0.71 (0.08) | 0.69 (0.10) | 0.88 (0.16)
  Month 36 Limited Cognitive Capacity (n=34,21,8) | 0.67 (0.08) | 0.73 (0.10) | 0.85 (0.17)
  Month 36 Cardiac and Renal Dysfunction (n=33,21,8) | 0.58 (0.08) | 0.57 (0.10) | 0.76 (0.16)
  Month 36 SE of Corticosteroids (n=33,21,8) | 0.44 (0.09) | 0.39 (0.11) | 0.58 (0.18)
  Month 36 IGGH (n=33,20,8) | 0.54 (0.08) | 0.33 (0.10) | 0.23 (0.15)
  Month 36 TAPD (n=34,21,8) | 0.77 (0.09) | 0.82 (0.11) | 0.68 (0.18)
  Month 36 Global Score (n=33,21,8) | 0.64 (0.06) | 0.63 (0.08) | 0.70 (0.12)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Limited Physical Capacity; Test type: Superiority or Other; p = 0.3093, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.10 to 0.33], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Limited Physical Capacity; Test type: Superiority or Other; p = 0.3223, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.12 to 0.36], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Limited Cognitive Capacity; Test type: Superiority or Other; p = 0.4858, Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.14 to 0.30], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Limited Cognitive Capacity; Test type: Superiority or Other; p = 0.3679, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.13 to 0.36], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Cardiac and Renal Dysfunction; Test type: Superiority or Other; p = 0.6416, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.27 to 0.17], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Cardiac and Renal Dysfunction; Test type: Superiority or Other; p = 0.4241, Mixed Models Analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.34 to 0.14], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Side Effects of Corticosteroids; Test type: Superiority or Other; p = 0.2133, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.09 to 0.39], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Side Effects of Corticosteroids; Test type: Superiority or Other; p = 0.1918, Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.09 to 0.44], Standard Error of Mean 0.13
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Increased Growth of Gum and Hair; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.55 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Increased Growth of Gum and Hair; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.59 to -0.13], Standard Error of Mean 0.12
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Transplantation-Associated Psychological Distress; Test type: Superiority or Other; p = 0.2012, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.08 to 0.40], Standard Error of Mean 0.12
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Transplantation-Associated Psychological Distress; Test type: Superiority or Other; p = 0.8986, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.25 to 0.29], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Global Score; Test type: Superiority or Other; p = 0.6724, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.13 to 0.20], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Global Score; Test type: Superiority or Other; p = 0.9297, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.18 to 0.19], Standard Error of Mean 0.09
Statistical Analysis 15: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Limited Physical Capacity; Test type: Superiority or Other; p = 0.8682, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.28 to 0.23], Standard Error of Mean 0.13
Statistical Analysis 16: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Limited Physical Capacity; Test type: Superiority or Other; p = 0.3392, Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.18 to 0.53], Standard Error of Mean 0.18
Statistical Analysis 17: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Limited Cognitive Capacity; Test type: Superiority or Other; p = 0.6545, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.20 to 0.32], Standard Error of Mean 0.13
Statistical Analysis 18: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Limited Cognitive Capacity; Test type: Superiority or Other; p = 0.3253, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.18 to 0.55], Standard Error of Mean 0.19
Statistical Analysis 19: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Cardiac and Renal Dysfunction; Test type: Superiority or Other; p = 0.9698, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.26 to 0.25], Standard Error of Mean 0.13
Statistical Analysis 20: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Cardiac and Renal Dysfunction; Test type: Superiority or Other; p = 0.3065, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.17 to 0.54], Standard Error of Mean 0.18
Statistical Analysis 21: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Side Effects of Corticosteroids; Test type: Superiority or Other; p = 0.7147, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.33 to 0.23], Standard Error of Mean 0.14
Statistical Analysis 22: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Side Effects of Corticosteroids; Test type: Superiority or Other; p = 0.4852, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.25 to 0.53], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Increased Growth of Gum and Hair; Test type: Superiority or Other; p = 0.0888, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.46 to 0.03], Standard Error of Mean 0.13
Statistical Analysis 24: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Increased Growth of Gum and Hair; Test type: Superiority or Other; p = 0.0719, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.65 to 0.03], Standard Error of Mean 0.17
Statistical Analysis 25: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Transplantation-Associated Psychological Distress; Test type: Superiority or Other; p = 0.7531, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.24 to 0.33], Standard Error of Mean 0.14
Statistical Analysis 26: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Transplantation-Associated Psychological Distress; Test type: Superiority or Other; p = 0.6412, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.49 to 0.30], Standard Error of Mean 0.20
Statistical Analysis 27: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Global Score; Test type: Superiority or Other; p = 0.9186, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.20 to 0.18], Standard Error of Mean 0.10
Statistical Analysis 28: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Global Score; Test type: Superiority or Other; p = 0.6629, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.21 to 0.33], Standard Error of Mean 0.14

26. Secondary Outcome: Least Squares Means of Severity of Dyspepsia Assessment (SODA) Subscales at Months 24 & 36
Description: SODA:17-item health scale, assessed participant-reported perceptions of dyspepsia; consists of 3 subscales: Pain Intensity (PI, 6-items to assess pain and intensity of abdominal discomfort; Range: 2 to 47, higher score indicates greater pain and abdominal discomfort), Non-Pain Symptoms (NPS, 7-items to assess severity and impact of non-pain symptoms: burping/belching, heartburn, bloating, flatulence, sour taste, nausea, and bad breath; Range: 7 to 35, higher scores indicate increased symptom severity and influence), and Satisfaction (4-items to assess degree of satisfaction with abdominal discomfort; Range: 2 to 23, higher scores indicate more satisfaction).
  Model contained treatment, visit and treatment by visit interaction as fixed effects and Baseline (predose in Study A3921030) as a covariate. A first-order autoregressive variance-covariance structure was used.
Time Frame: Months 24, 36
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 49 | 41 | 25
Score
  Month 24 PI Total Converted Score (n=46,39,24) | 9.51 (1.16) | 7.66 (1.26) | 10.73 (1.59)
  Month 24 NPS Converted Score | 11.44 (0.42) | 11.24 (0.46) | 12.25 (0.58)
  Month 24 Satisfaction Converted Score (n=49,41,24) | 17.22 (0.66) | 18.11 (0.72) | 16.33 (0.94)
  Month 36 PI Total Converted Score (n=40,27,10) | 9.63 (1.25) | 8.03 (1.51) | 10.59 (2.45)
  Month 36 NPS Converted Score (n=42,28,10) | 11.31 (0.45) | 11.14 (0.55) | 12.44 (0.91)
  Month 36 Satisfaction Converted Score (n=42,28,10) | 17.44 (0.72) | 17.90 (0.87) | 16.31 (1.45)
Statistical Analysis 1: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Pain Intensity Total Converted Score; Test type: Superiority or Other; p = 0.2826, Mixed Models Analysis; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-5.22 to 1.53], Standard Error of Mean 1.72
Statistical Analysis 2: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Pain Intensity Total Converted Score; Test type: Superiority or Other; p = 0.5371, Mixed Models Analysis; Mean Difference (Final Values) = 1.22, 95% CI 2-sided [-2.65 to 5.09], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Non-Pain Symptoms Converted Score; Test type: Superiority or Other; p = 0.7503, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-1.41 to 1.02], Standard Error of Mean 0.62
Statistical Analysis 4: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Non-Pain Symptoms Converted Score; Test type: Superiority or Other; p = 0.2610, Mixed Models Analysis; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.60 to 2.21], Standard Error of Mean 0.72
Statistical Analysis 5: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 24 Satisfaction Converted Score; Test type: Superiority or Other; p = 0.3656, Mixed Models Analysis; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-1.04 to 2.82], Standard Error of Mean 0.98
Statistical Analysis 6: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 24 Satisfaction Converted Score; Test type: Superiority or Other; p = 0.4405, Mixed Models Analysis; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-3.16 to 1.37], Standard Error of Mean 1.15
Statistical Analysis 7: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Pain Intensity Total Converted Score; Test type: Superiority or Other; p = 0.4135, Mixed Models Analysis; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-5.45 to 2.25], Standard Error of Mean 1.96
Statistical Analysis 8: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Pain Intensity Total Converted Score; Test type: Superiority or Other; p = 0.7272, Mixed Models Analysis; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-4.45 to 6.37], Standard Error of Mean 2.75
Statistical Analysis 9: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Non-Pain symptoms Converted Score; Test type: Superiority or Other; p = 0.8111, Mixed Models Analysis; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-1.56 to 1.22], Standard Error of Mean 0.71
Statistical Analysis 10: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Non-Pain Symptoms Converted Score; Test type: Superiority or Other; p = 0.2636, Mixed Models Analysis; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-0.86 to 3.13], Standard Error of Mean 1.02
Statistical Analysis 11: Comparison: Cyclosporine vs Tofacitinib Less Intensive (LI); Month 36 Satisfaction Converted Score; Test type: Superiority or Other; p = 0.6890, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-1.77 to 2.67], Standard Error of Mean 1.13
Statistical Analysis 12: Comparison: Cyclosporine vs Tofacitinib More Intensive (MI); Month 36 Satisfaction Converted Score; Test type: Superiority or Other; p = 0.4853, Mixed Models Analysis; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-4.31 to 2.05], Standard Error of Mean 1.62

27. Secondary Outcome: Mean Trough Levels of Tofacitinib by Visit
Description: The dates and times were recorded for the 6 doses of tofacitinib administered before each scheduled pharmacokinetic (PK) sampling. The participant was instructed to follow a 12 hourly schedule for these 6 doses of tofacitinib, with each dose administered within 1 hour of the scheduled time. Trough samples were collected 0 to 10 minutes prior to the morning dose. 1 hour postdose samples were required within 10 minutes of the nominal time point. Samples taken at -2 hours predose and at time points >1 hour post dose were required within 30 minutes of the nominal time point.
Time Frame: Months 18 and 24 (-2 hours, predose, 1 hour, 2 hours), Month 30 (predose, 1 hour and 2 hours), Month 36 (predose, 1, 2, and 4 hours), Months 42, 48, 54, 60, 66, 72 (predose and 2 hours)
Population: Safety Analysis Set. n is the number of participants with the assessment at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Number analyzed (Participants) | 58 | 46
ng/mL
  Month 18 Predose -2 hours (n=31,22) | 13.20 (10.43) | 10.68 (6.86)
  Month 18 Predose | 12.45 (11.83) | 15.27 (24.14)
  Month 18 1 hour (n=58,45) | 56.62 (32.96) | 56.58 (37.56)
  Month 18 2 hours (n=26,23) | 59.55 (25.87) | 56.60 (28.85)
  Month 24 Predose -2 hours (n=18,15) | 11.71 (11.77) | 8.95 (8.72)
  Month 24 Predose (n=50,32) | 9.93 (14.50) | 7.42 (4.88)
  Month 24 1 hour (n=49,31) | 44.06 (26.16) | 41.93 (27.27)
  Month 24 2 hours (n=28,15) | 37.73 (14.00) | 34.15 (15.27)
  Month 30 Predose (n=35,21) | 8.70 (8.53) | 6.89 (6.94)
  Month 30 1 hour (n=35,21) | 39.15 (16.06) | 44.12 (19.99)
  Month 30 2 hours (n=34,19) | 38.07 (11.42) | 37.16 (17.51)
  Month 36 Predose (n=31,15) | 6.35 (4.68) | 8.33 (10.76)
  Month 36 1 hour (n=30,14) | 46.09 (12.54) | 38.07 (14.06)
  Month 36 2 hours (n=30,15) | 38.11 (14.41) | 31.76 (7.45)
  Month 36 4 hours (n=30,15) | 24.03 (10.34) | 21.46 (4.33)
  Month 42 Predose (n=31,14) | 11.42 (12.07) | 7.00 (5.34)
  Month 42 2 hours (n=30,12) | 35.27 (15.57) | 34.33 (11.10)
  Month 48 Predose (n=32,14) | 7.58 (6.94) | 13.78 (11.05)
  Month 48 2 hours (n=32,12) | 38.46 (12.36) | 41.10 (12.35)
  Month 54 Predose (n=30,11) | 7.86 (5.52) | 7.09 (6.45)
  Month 54 2 hours (n=30,10) | 41.18 (12.25) | 48.03 (10.39)
  Month 60 Predose (n=23,10) | 6.58 (3.82) | 7.31 (5.41)
  Month 60 2 hours (n=23,10) | 39.43 (9.26) | 38.98 (13.33)
  Month 66 Predose (n=22,10) | 7.53 (9.19) | 5.81 (6.03)
  Month 66 2 hours (n=21,10) | 36.17 (12.74) | 41.12 (12.27)
  Month 72 Predose (n=16,8) | 8.30 (7.22) | 5.37 (5.05)
  Month 72 2 hours (n=16,8) | 38.55 (14.38) | 38.93 (13.19)

28. Secondary Outcome: Mean Trough Levels of Cyclosporine by Visit
Description: All CsA samples were taken predose (collected 0 to 10 minutes prior to the morning dose).
Time Frame: Predose: Months 18, 24, 36, 48, 60, 72
Population: Safety Analysis Set. n is the number of participants with the assessment at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cyclosporine
Number analyzed (Participants) | 58
ng/mL
  Month 18 | 113.88 (98.73)
  Month 24 (n=54) | 89.52 (45.23)
  Month 36 (n=50) | 101.10 (100.63)
  Month 48 (n=39) | 88.54 (62.45)
  Month 60 (n=35) | 95.00 (115.74)
  Month 72 (n=23) | 135.30 (188.05)

ADVERSE EVENTS:
Time Frame: Adverse events (serious and non-serious) were recorded on the Case Report Form from the time the subject had taken at least 1 dose of study treatment through the follow-up visit at Month 74 or 2 months following discontinuation of treatment.
Description: The same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Cyclosporine | Tofacitinib Less Intensive (LI) | Tofacitinib More Intensive (MI)
Serious Adverse Events (participants affected / at risk) | 40/64 | 32/60 | 31/54
Other Adverse Events (participants affected / at risk) | 49/64 | 55/60 | 45/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=64) | Tofacitinib Less Intensive (LI) (N=60) | Tofacitinib More Intensive (MI) (N=54)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperparathyrodism (Endocrine disorders) | 0 | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 3 | 0 | 1
Drug ineffective (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 2 | 3 | 2
Transplant rejection (Immune system disorders) | 6 | 2 | 1
Abscess (Infections and infestations) | 0 | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Aspergilloma (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1
Gas gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 2 | 0
H1N1 influenza (Infections and infestations) | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 2 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 2
Mycobacterium chelonae infection (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 3 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 3
Sinusitis (Infections and infestations) | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Exposure via father (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 2
Liver function test abnormal (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Brain mass (Nervous system disorders) | 0 | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Renal injury (Renal and urinary disorders) | 1 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cyclosporine (N=64) | Tofacitinib Less Intensive (LI) (N=60) | Tofacitinib More Intensive (MI) (N=54)
Hypertension (Vascular disorders) | 6 | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 8 | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 4 | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 1
Constipation (Gastrointestinal disorders) | 4 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 4
Nausea (Gastrointestinal disorders) | 6 | 7 | 2
Vomiting (Gastrointestinal disorders) | 9 | 8 | 2
Chest pain (General disorders) | 7 | 2 | 1
Fatigue (General disorders) | 3 | 5 | 5
Oedema peripheral (General disorders) | 4 | 10 | 4
Peripheral swelling (General disorders) | 3 | 6 | 0
Pyrexia (General disorders) | 3 | 7 | 3
Transplant rejection (Immune system disorders) | 5 | 1 | 0
BK virus infection (Infections and infestations) | 0 | 6 | 1
Bronchitis (Infections and infestations) | 4 | 4 | 1
Epstein-Barr viraemia (Infections and infestations) | 1 | 1 | 3
Fungal skin infection (Infections and infestations) | 0 | 1 | 3
Gastroenteritis (Infections and infestations) | 2 | 6 | 2
Herpes zoster (Infections and infestations) | 3 | 11 | 5
Nasopharyngitis (Infections and infestations) | 5 | 4 | 3
Onychomycosis (Infections and infestations) | 2 | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 10 | 13
Urinary tract infection (Infections and infestations) | 4 | 4 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 4 | 6
Blood creatine phosphokinase increased (Investigations) | 3 | 4 | 5
Blood creatinine increased (Investigations) | 7 | 1 | 2
Cardiac murmur (Investigations) | 2 | 4 | 4
Weight decreased (Investigations) | 2 | 5 | 0
Weight increased (Investigations) | 4 | 5 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 2
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 8 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 1
Dizziness (Nervous system disorders) | 4 | 2 | 2
Headache (Nervous system disorders) | 8 | 7 | 3
Tremor (Nervous system disorders) | 1 | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 5 | 4
Depression (Psychiatric disorders) | 2 | 4 | 0
Insomnia (Psychiatric disorders) | 6 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 5 | 1
Proteinuria (Renal and urinary disorders) | 4 | 4 | 3
Menorrhagia (Reproductive system and breast disorders) | 0/20 | 1/19 | 1/14
Vulval disorder (Reproductive system and breast disorders) | 0/20 | 1/19 | 0/14
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6 | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 2/20 | 0/19 | 0/14
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 4
Postmenopause (Social circumstances) | 0/20 | 0/19 | 1/14
Haematoma (Vascular disorders) | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less